CLINICAL TRIAL: NCT03737110
Title: Phase 3, Double-Blind, Placebo-Controlled, Randomized Withdrawal Study With Open-label Extension, to Assess the Efficacy and Safety of Rilonacept Treatment in Subjects With Recurrent Pericarditis
Brief Title: Study to Assess the Efficacy and Safety of Rilonacept Treatment in Participants With Recurrent Pericarditis
Acronym: RHAPSODY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kiniksa Pharmaceuticals (UK), Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kiniksa Pharmaceuticals International, plc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KPL-914-C002; 2018-002719-87 (EudraCT Number)
Record Dates: First submitted 2018-10-30; First posted 2018-11-09 (Actual); Results first posted 2021-07-13 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Recurrent Pericarditis
MeSH Terms: conditions — Pericarditis | interventions — rilonacept

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rilonacept (Experimental): RI period: single-blind rilonacept 320 mg (or 4.4 mg/kg in pediatric participants) SC, followed by 160 mg (or 2.2 mg/kg in pediatric participants) injections once weekly.
  RW period: eligible participants randomized to double-blinded administration of rilonacept 160 mg (or 2.2 mg/kg in pediatric participants) SC injections once weekly. Participants with pericarditis recurrence who meet the protocol criteria for bailout rilonacept (report at least 1 day with pericarditis pain ≥4 on the 11-point NRS and have 1 CRP value ≥ 1 mg/dL [either on the same day or separated by no more than 7 days]) receive bailout rilonacept (2 open-label injections of 160 mg rilonacept [or 4.4 mg/kg for pediatric participants]) irrespective of randomized treatment assignment and as soon as at least 5 days have passed since the last study drug injection.
  LTE period: open-label administration of rilonacept 160 mg (or 2.2 mg/kg in pediatric participants) SC injections once weekly.
  Interventions: Drug: Rilonacept
- Placebo (Placebo Comparator): RI period: single-blind rilonacept 320 mg (or 4.4 mg/kg in pediatric participants) SC, followed by 160 mg (or 2.2 mg/kg in pediatric participants) injections once weekly.
  RW period: eligible participants randomized to placebo SC injections once weekly. Participants with pericarditis recurrence who meet the protocol criteria for bailout rilonacept (report at least 1 day with pericarditis pain ≥4 on the 11-point NRS and have 1 CRP value ≥ 1 mg/dL [either on the same day or separated by no more than 7 days]) receive bailout rilonacept (2 open-label injections of 160 mg rilonacept [or 4.4 mg/kg for pediatric participants]) irrespective of randomized treatment assignment and as soon as at least 5 days have passed since the last study drug injection.
  LTE period: open-label administration of rilonacept 160 mg (or 2.2 mg/kg in pediatric participants) SC injections once weekly.
  Interventions: Drug: Rilonacept; Drug: Placebo

INTERVENTIONS:
Drug: Rilonacept — Rilonacept 320 mg (or 4.4 mg/kg in pediatric participants ≥12 and <18 years old) SC , followed by 160 mg (or 2.2 mg/kg in pediatric participants ≥12 and <18 years old) injections once weekly
  Other Names: KPL-914; Arcalyst® for Cryopyrin-Associated Periodic Syndromes (CAPS)
Drug: Placebo — Placebo SC injections once weekly
  Arms: Placebo

SUMMARY:
The primary objective of this study was to assess the efficacy of rilonacept treatment in participants with recurrent pericarditis.

DETAILED DESCRIPTION:
In the single-blind run-in (RI) period, rilonacept 320 mg (or 4.4 mg/kg in pediatric participants ≥12 and <18 years old) subcutaneous (SC), followed by 160 mg (or 2.2 mg/kg in pediatric participants ≥12 and <18 years old) injections once weekly.

During the Randomized-Withdrawal (RW) period, eligible participants are randomized 1:1 to double-blinded administration of study drug:

* Rilonacept 160 mg (or 2.2 mg/kg in pediatric participants ≥12 and <18 years old) SC injections once weekly
* Matching placebo SC injections once weekly.

Participants with pericarditis recurrence who meet the protocol criteria for bailout rilonacept (report at least 1 day with pericarditis pain ≥4 on the 11-point numerical rating scale (NRS) and have 1 C-reactive protein (CRP) value ≥ 1 mg/dL [either on the same day or separated by no more than 7 days]) receive bailout rilonacept (2 open-label injections of 160 mg rilonacept [or 4.4 mg/kg for pediatric subjects]) irrespective of randomized treatment assignment and as soon as at least 5 days have passed since the last study drug injection.

Upon completion of the RW period (i.e., when the prespecified number of primary efficacy endpoints [clinical events committee-confirmed pericarditis recurrence] events have occurred), all participants who did not discontinue study drug have an option to continue treatment with open-label rilonacept in the Long-Term Extension (LTE) or to withdraw from the study. Participants still in the RI period at the time that the RW period has ended and the LTE is opened will have the option to enter the LTE directly when they have completed the RI period and have met the definition of clinical response or to withdraw from the study.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female aged 12 or older
2. Has a diagnosis of recurrent pericarditis
3. Must provide Informed Consent
4. Presents with at least the third episode of pericarditis during screening.
5. Has received nonsteroidal anti-inflammatory drugs (NSAIDs) and/or colchicine and/or corticosteroids (in any combination), if used, at stable dose levels (or at least not increased) for at least 3 days prior to first study drug administration
6. Female subjects must be postmenopausal, or incapable of pregnancy or permanently sterile, or if of childbearing potential must agree to use highly-effective method of contraception.
7. Must be up-to-date with all immunizations, in agreement with current local immunization guidelines for immunosuppressed subjects, before first study drug administration.
8. Is able to adequately maintain a daily subject diary according to protocol.
9. Agrees to refrain from making any new, major lifestyle changes that may affect pericarditis symptoms (e.g., changing exercise pattern) from the time that the informed consent form (ICF) is signed through the end of the double-blind randomized withdrawal period.

Key Exclusion Criteria:

1. Has a diagnosis of pericarditis that is secondary to specific prohibited etiologies.
2. Has a history of immunosuppression, including positive human immunodeficiency virus (HIV) test results.
3. Has a history of myeloproliferative disorder.
4. Has a history of demyelinating disease or symptoms suggestive of multiple sclerosis.
5. Has a history of active or latent tuberculosis (TB) prior to screening
6. Has chest x-ray at screening or within 12 weeks before receiving first administration of study drug, with evidence of malignancy or abnormality consistent with prior or active TB infection.
7. Has a history of positive or intermediate results for hepatitis B surface antigen, hepatitis B core antibody, or hepatitis C virus antibody at screening.
8. Has a history of malignancy of any organ system within the past 5 years before screening (other than a successfully treated non metastatic cutaneous squamous cell carcinoma or basal cell carcinoma and/or localized carcinoma in situ of the cervix).
9. Has a known or suspected current active infection or a history of chronic or recurrent infectious disease, including, but not limited to, chronic renal infection, chronic chest infection, sinusitis, recurrent urinary tract infection, or an open, draining infected skin wound.
10. Has had an organ transplant.
11. In the Investigator's opinion, has a history of alcoholism or drug/chemical abuse within 2 years before screening.
12. Has a known hypersensitivity to rilonacept or to any of its excipients.
13. Has received an investigational drug during the 30 days before screening or is planning to receive an investigational drug (other than that administered during this study) or use an investigational device at any time during the study.
14. In the Investigator's opinion, has any other medical condition that could adversely affect the subject's participation or interfere with study evaluations.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-05-29 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations Study Director, Study Director — Kiniksa Pharmaceuticals (UK), Ltd.
Locations (21):
- United States (12):
  - Cedars-Sinai Medical Institute, Los Angeles, California
  - Arthritis and Rheumatology of Georgia, Atlanta, Georgia
  - The Loretto Hospital, Chicago, Illinois
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic - PPDS, Rochester, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Cardiology Consultants of Philadelphia, Yardley, Pennsylvania
  - Intermountain Healthcare, Murray, Utah
  - University Of Vermont Medical Center, Burlington, Vermont
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
- Australia (2):
  - HeartCare Partners Clinical Research Unit, Milton, Queensland
  - GenesisCare - Cardiology Research, Doncaster East, Victoria
- Israel (4):
  - Bnai Zion Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Galilee Medical Center, Nahariya
  - Sheba Medical Center at Tel-Hashomer, Ramat Gan
- Italy (3):
  - Ospedale Pediatrico Bambino Gesù, Rome, Lazio
  - ASST Fatebenefratelli Sacco - Ospedale Fatebenefratelli e Oftalmico, Milan, Lombardy
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Piedmont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klein AL, Imazio M, Cremer P, Brucato A, Abbate A, Fang F, Insalaco A, LeWinter M, Lewis BS, Lin D, Luis SA, Nicholls SJ, Pano A, Wheeler A, Paolini JF; RHAPSODY Investigators. Phase 3 Trial of Interleukin-1 Trap Rilonacept in Recurrent Pericarditis. N Engl J Med. 2021 Jan 7;384(1):31-41. doi: 10.1056/NEJMoa2027892. Epub 2020 Nov 16. PMID 33200890
- [Derived] Cremer PC, Lin D, Luis SA, Petersen J, Abbate A, Jellis CL, Kwon D, Brucato A, Fang F, Insalaco A, LeWinter M, Lewis BS, Zou L, Nicholls SJ, Klein AL, Imazio M, Paolini JF; RHAPSODY Investigators. Pericardial late gadolinium enhancement and time to recurrence: a substudy from RHAPSODY, a phase 3 clinical trial of rilonacept in recurrent pericarditis. Eur Heart J Imaging Methods Pract. 2023 May 26;1(1):qyad003. doi: 10.1093/ehjimp/qyad003. eCollection 2023 May. PMID 39044797
- [Derived] Brucato A, Trotta L, Arad M, Cremer PC, Insalaco A, Klutstein M, LeWinter M, Lin D, Luis SA, Wasserstrum Y, Clair J, Wang S, Klein AL, Imazio M, Paolini JF; RHAPSODY Investigators. Absence of Pericarditis Recurrence in Rilonacept-Treated Patients With COVID-19 and SARS-CoV-2 Vaccination: Results From the RHAPSODY Long-term Extension. CJC Open. 2024 Mar 4;6(6):805-810. doi: 10.1016/j.cjco.2024.02.002. eCollection 2024 Jun. PMID 39022168
- [Derived] Imazio M, Klein AL, Brucato A, Abbate A, Arad M, Cremer PC, Insalaco A, LeWinter MM, Lewis BS, Lin D, Luis SA, Nicholls SJ, Sutej P, Wasserstrum Y, Clair J, Agarwal I, Wang S, Paolini JF; RHAPSODY Investigators. Sustained Pericarditis Recurrence Risk Reduction With Long-Term Rilonacept. J Am Heart Assoc. 2024 Mar 19;13(6):e032516. doi: 10.1161/JAHA.123.032516. Epub 2024 Mar 12. PMID 38471825
- [Derived] Thomas GK, Bonaventura A, Vecchie A, van Tassell B, Imazio M, Klein A, Luis SA, Abbate A. Interleukin-1 Blockers for the Treatment of Recurrent Pericarditis: Pathophysiology, Patient-Reported Outcomes, and Perspectives. J Cardiovasc Pharmacol. 2024 Jun 1;83(6):503-510. doi: 10.1097/FJC.0000000000001435. PMID 37163222
- [Derived] Brucato A, Wheeler A, Luis SA, Abbate A, Cremer PC, Zou L, Insalaco A, Lewinter M, Lewis BS, Lin D, Nicholls S, Pancrazi M, Klein AL, Imazio M, Paolini JF. Transition to rilonacept monotherapy from oral therapies in patients with recurrent pericarditis. Heart. 2023 Jan 27;109(4):297-304. doi: 10.1136/heartjnl-2022-321328. PMID 36316102
- [Derived] Brucato A, Lim-Watson MZ, Klein A, Imazio M, Cella D, Cremer P, LeWinter MM, Luis SA, Lin D, Lotan D, Pancrazi M, Trotta L, Klooster B, Litcher-Kelly L, Zou L, Magestro M, Wheeler A, Paolini JF; RHAPSODY Investigators. Interleukin-1 Trap Rilonacept Improved Health-Related Quality of Life and Sleep in Patients With Recurrent Pericarditis: Results From the Phase 3 Clinical Trial RHAPSODY. J Am Heart Assoc. 2022 Oct 18;11(20):e023252. doi: 10.1161/JAHA.121.023252. Epub 2022 Oct 17. PMID 36250662
- [Derived] Klein AL, Imazio M, Brucato A, Cremer P, LeWinter M, Abbate A, Lin D, Martini A, Beutler A, Chang S, Fang F, Gervais A, Perrin R, Paolini JF. RHAPSODY: Rationale for and design of a pivotal Phase 3 trial to assess efficacy and safety of rilonacept, an interleukin-1alpha and interleukin-1beta trap, in patients with recurrent pericarditis. Am Heart J. 2020 Oct;228:81-90. doi: 10.1016/j.ahj.2020.07.004. Epub 2020 Jul 14. PMID 32866928

RESULTS

PARTICIPANT FLOW:
Groups:
- Run-in Period: Single-blind rilonacept 320 mg (or 4.4 mg/kg in pediatric participants ≥ 12 and < 18 years old) subcutaneous (SC), followed by 160 mg (or 2.2 mg/kg in pediatric participants ≥12 and <18 years old) injections once weekly for 12 weeks.
  Participants still in the Run-in Period at the time that the Randomized Withdrawal Period has ended (ie, when the prespecified number of primary efficacy endpoint events have occurred) and the Long-Term Extension (LTE) Period is opened will have the option to enter the LTE directly when they have completed the RI period and have met the definition of clinical response or to withdraw from the study.
- Randomized Withdrawal Period: Rilonacept: Double-blind rilonacept 160 mg (or 2.2 mg/kg in pediatric participants ≥ 12 and < 18 years old) SC injections once weekly.
  Participants with pericarditis recurrence who meet the protocol criteria for bailout rilonacept (report at least 1 day with pericarditis pain ≥4 on the 11-point numerical rating scale (NRS) and have 1 C-reactive protein (CRP) value ≥ 1 mg/dL [either on the same day or separated by no more than 7 days]) receive bailout rilonacept (2 open-label injections of 160 mg rilonacept [or 4.4 mg/kg for pediatric participants]) irrespective of randomized treatment assignment and as soon as at least 5 days have passed since the last study drug injection.
  Upon completion of the RW period (ie, when the prespecified number of primary efficacy endpoint events has occurred), all participants who did not discontinue study drug have an option to continue treatment with open-label rilonacept in the LTE period or to withdraw from the study.
- Randomized Withdrawal Period: Placebo: Double-blind placebo SC injections once weekly.
  Participants with pericarditis recurrence who meet the protocol criteria for bailout rilonacept (report at least 1 day with pericarditis pain ≥4 on the 11-point NRS and have 1 CRP value ≥ 1 mg/dL [either on the same day or separated by no more than 7 days]) receive bailout rilonacept (2 open-label injections of 160 mg rilonacept [or 4.4 mg/kg for pediatric participants]) irrespective of randomized treatment assignment and as soon as at least 5 days have passed since the last study drug injection.
  Upon completion of the RW period (ie, when the prespecified number of primary efficacy endpoint events has occurred), all participants who did not discontinue study drug have an option to continue treatment with open-label rilonacept in the LTE period or to withdraw from the study.
- Long Term Extension: Non-Randomized: Participants who entered the LTE directly from RI after protocol-specified 22 adjudicated pericarditis recurrence events had accrued received up to 24 months of open-label rilonacept 160 mg (or 2.2 mg/kg for pediatric participants) SC injections once weekly based on their clinical status and at the discretion of the Investigator.
- Long Term Extension: Randomized, Recurrence (RW): Participants with recurrence as evaluated based on CEC adjudication in Randomization Withdrawal period received up to 24 months of open-label rilonacept 160 mg (or 2.2 mg/kg for pediatric participants) SC injections once weekly based on their clinical status and at the discretion of the Investigator.
- Long Term Extension: Randomized, No Recurrence (RW): Participants with no recurrence as evaluated based on CEC adjudication in Randomization Withdrawal period received up to 24 months of open-label rilonacept 160 mg (or 2.2 mg/kg for pediatric participants) SC injections once weekly based on their clinical status and at the discretion of the Investigator.
Period: Run-in (RI) Period
Arm/Group | Run-in Period | Randomized Withdrawal Period: Rilonacept | Randomized Withdrawal Period: Placebo | Long Term Extension: Non-Randomized | Long Term Extension: Randomized, Recurrence (RW) | Long Term Extension: Randomized, No Recurrence (RW)
Started | 86 | 0 | 0 | 0 | 0 | 0
Continue to RW Period | 61 | 0 | 0 | 0 | 0 | 0
Continue Directly to LTE Period | 15 | 0 | 0 | 0 | 0 | 0
Completed | 76 | 0 | 0 | 0 | 0 | 0
Not Completed | 10 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Did Not Meet Clinical Response Criteria | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0 | 0 | 0 | 0
Period: Randomized Withdrawal (RW) Period
Arm/Group | Run-in Period | Randomized Withdrawal Period: Rilonacept | Randomized Withdrawal Period: Placebo | Long Term Extension: Non-Randomized | Long Term Extension: Randomized, Recurrence (RW) | Long Term Extension: Randomized, No Recurrence (RW)
Started (Met protocol-defined clinical response criteria and entered into RW Period.) | 0 | 30 | 31 | 0 | 0 | 0
Completed (Completed, Continuing into LTE) | 0 | 29 | 30 | 0 | 0 | 0
Not Completed | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Completed, Not Continuing into LTE | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0
Period: Long-Term Extension (LTE) Period
Arm/Group | Run-in Period | Randomized Withdrawal Period: Rilonacept | Randomized Withdrawal Period: Placebo | Long Term Extension: Non-Randomized | Long Term Extension: Randomized, Recurrence (RW) | Long Term Extension: Randomized, No Recurrence (RW)
Started | 0 (Participants who entered the LTE directly from RI after protocol-specified 22 adjudicated pericarditis recurrence events had accrued.) | 0 (1 participant withdrew consent prior to entering LTE.) | 0 | 15 | 25 | 34
Completed | 0 | 0 | 0 | 13 | 24 | 32
Not Completed | 0 | 0 | 0 | 2 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Investigator Decision due to Serious Adverse Event | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants entering the double-blind Randomized Withdrawal Treatment Period.
Groups:
- Randomized Withdrawal Period: Rilonacept: Double-blind rilonacept 160 mg (or 2.2 mg/kg in pediatric participants ≥ 12 and < 18 years old) SC injections once weekly.
- Randomized Withdrawal Period: Placebo: Double-blind placebo SC injections once weekly.
- Total: Total of all reporting groups
Arm/Group | Randomized Withdrawal Period: Rilonacept | Randomized Withdrawal Period: Placebo | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (15.70) | 44.8 (14.47) | 46.4 (15.05)
Age, Customized [Count of Participants; unit: Participants]
  12 to 17 years | 1 | 2 | 3
  18 to 64 years | 24 | 27 | 51
  65 to 78 years | 5 | 2 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 14 | 15 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 30 | 31 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 28 | 28 | 56
  Black or African American | 1 | 3 | 4
  Other, Not Specified | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Pericarditis Recurrence in the RW Period
Description: Time to pericarditis recurrence (from randomization to 1st recurrence). Kaplan-Meier. Clinical Events Committee (CEC)-confirmed recurrences used for primary analysis. Recurrence defined as recurrence typical pericarditis pain with supportive objective evidence. CEC-adjudicated recurrences defined as:1) Re-appearance/worsening pericarditis pain (1 NRS ≥ 4) AND elevated CRP (≥1.0 mg/dL) on same day/separated by ≤ 7 days OR 2) Re-appearance/worsening pericarditis pain (1 NRS ≥ 4) AND abnormal CRP (> 0.5 mg/dL) on same day/separated by ≤ 7 days AND 1 supportive evidence OR 3) Re-appearance/worsening pericarditis pain (no NRS ≥ 4) AND elevated CRP (≥ 1.0 mg/dL) not attributable to other causes AND 1 supportive evidence. Supportive evidence: White blood cell count > upper limit normal, fever > 38C, pericardial rub, electrocardiogram changes consistent with pericarditis, new/worsening pericardial effusion (echocardiogram), new/worsening pericardial inflammation (magnetic resonance imaging).
Time Frame: RW Period (mean 24.8 weeks)
Population: Intent-to-Treat (ITT) Analysis Set: all participants who were randomized in the RW period.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Randomized Withdrawal Period: Rilonacept | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 30 | 31
weeks | NA [NA to NA] — The median was not reached due to low number of participants with an event at data cutoff. | 8.6 [4.0 to 11.7]
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: Rilonacept vs Randomized Withdrawal Period: Placebo; Test type: Superiority; p < 0.0001, Log Rank — Two-sided p-value is from the log-rank test stratified by oral corticosteroid use at Run-In Baseline; Hazard Ratio (HR) = 0.04, 95% CI 2-sided [0.01 to 0.18] — Calculated based on a Cox proportional-hazards model with treatment as covariate and stratified by oral corticosteroid use at run-in baseline

2. Secondary Outcome: Major Secondary Efficacy Endpoint: Percentage of Participants Who Maintained Clinical Response at Week 16 of the RW Period
Description: Participants were asked to select the score that best describes their average level of pericarditis pain over the previous 24 hours using an 11-point numerical rating scale (NRS), where zero (0) indicates 'no pain' and ten (10) indicates 'pain as bad as it could be'. Clinical response was defined as a weekly average of daily pericarditis pain on the NRS ≤ 2.0 and C-reactive protein (CRP) level ≤ 0.5 mg/dL, and on monotherapy of randomized study drug at Week 16.
Time Frame: RW Period Week 16
Population: ITT Week 16 Analysis Set: All participants randomized at least 16 weeks before data cutoff.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomized Withdrawal Period: Rilonacept | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 21 | 20
percentage of participants | 81.0 [58.1 to 94.6] | 20.0 [5.7 to 43.7]
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: Rilonacept vs Randomized Withdrawal Period: Placebo; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel — 95% confidence interval (CI) and p-value were analyzed using a Cochran-Mantel-Haenszel test adjusted by oral corticosteroid use and diagnosis of recurrent idiopathic pericarditis at run-in baseline; Odds Ratio (OR) = 12.727, 95% CI 2-sided [2.438 to 66.428]
Statistical Analysis 2: Comparison: Randomized Withdrawal Period: Rilonacept vs Randomized Withdrawal Period: Placebo; Test type: Superiority; Difference in percentages = 61.0, 95% CI 2-sided [36.7 to 85.2] — Differences between percentages are reported in percentage points. The 95% confidence intervals for the differences in percentages were based on a normal approximation

3. Secondary Outcome: Major Secondary Efficacy Endpoint: Percentage of Days With No or Minimal Pericarditis Pain at Week 16 of the RW Period
Description: Participants were asked to select the score that best describes their average level of pericarditis pain over the previous 24 hours using an 11-point numerical rating scale (NRS), where zero (0) indicates 'no pain' and ten (10) indicates 'pain as bad as it could be'. No or minimal pain was defined as non-missing NRS ≤ 2.
  The percentage of days with no or minimal pericarditis pain in the first 16 weeks was calculated for each participant using 16×7 as the denominator. Missing values in pain diary were counted as 0 day with no or minimal pain. Days of using oral rescue therapy or corticosteroid count as 0 day with no or minimal pain. If bailout rilonacept was used, each administration (loading dose or not) was counted as 7 days without qualifying no or minimal pain.
Time Frame: RW Period Week 16
Population: ITT Week 16 Analysis Set: All participants randomized at least 16 weeks before data cutoff.
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Randomized Withdrawal Period: Rilonacept | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 21 | 20
percentage of days | 98.6 (7.55) | 47.4 (7.26)
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: Rilonacept vs Randomized Withdrawal Period: Placebo; Test type: Superiority; p < 0.0001, ANCOVA — Two-sided p-value calculated using analysis of covariance with treatment, randomization strata and run-in baseline NRS weekly average category (NRS ≤ 2 versus NRS >2) as covariates; Least squares (LS) mean difference = 51.2, 95% CI 2-sided [34.5 to 68.0] — Least squares mean difference (rilonacept - placebo)

4. Secondary Outcome: Major Secondary Efficacy Endpoint: Percentage of Participants With Absent or Minimal Pericarditis Symptoms Based on the Patient Global Impression of Pericarditis Severity (PGIPS) at Week 16 of the RW Period
Description: Percentage of participants with no or minimal pericarditis symptoms at Week 16, based on the PGIPS, a single-item measure of the participant's impression of the overall severity of pericarditis symptoms at the time the questionnaire is administered using a 7-point rating scale ranging from absent (0=no recurrent pericarditis symptoms) to very severe (6=recurrent pericarditis symptoms that cannot be ignored and markedly limits daily activities).
  The exact 95% CI is calculated with randomization strata pooled. Participants who had received bailout rilonacept or rescue medication before the time point were considered nonresponders.
Time Frame: RW Period Week 16
Population: ITT Week 16 Analysis Set: All participants randomized at least 16 weeks before data cutoff.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomized Withdrawal Period: Rilonacept | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 21 | 20
percentage of participants | 81.0 [58.1 to 94.6] | 25.0 [8.7 to 49.1]
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: Rilonacept vs Randomized Withdrawal Period: Placebo; Test type: Superiority; p = 0.0006, Cochran-Mantel-Haenszel — 95% CI and p-value are analyzed using a Cochran-Mantel-Haenszel test adjusted by oral corticosteroid use and diagnosis of recurrent idiopathic pericarditis at RI baseline; Odds Ratio (OR) = 10.000, 95% CI 2-sided [2.136 to 46.826]
Statistical Analysis 2: Comparison: Randomized Withdrawal Period: Rilonacept vs Randomized Withdrawal Period: Placebo; Test type: Superiority; Difference in percentages = 56.0, 95% CI 2-sided [30.6 to 81.3] — [estimate comment as in outcome 2, analysis 2]

5. Secondary Outcome: Percentage of Participants Who Maintained Clinical Response at Week 24 of the RW Period
Description: Participants were asked to select the score that best describes their average level of pericarditis pain over the previous 24 hours using an 11-point numerical rating scale (NRS), where zero (0) indicates 'no pain' and ten (10) indicates 'pain as bad as it could be'. Clinical response was defined as a weekly average of daily pericarditis pain on the NRS ≤ 2.0 and C-reactive protein (CRP) level ≤ 0.5 mg/dL, and on monotherapy of randomized study drug at Week 24.
Time Frame: RW Period Week 24
Population: ITT Week 24 Analysis Set: All participants randomized at least 24 weeks before data cutoff.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomized Withdrawal Period: Rilonacept | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 17 | 15
percentage of participants | 76.5 [50.1 to 93.2] | 20.0 [4.3 to 48.1]
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: Rilonacept vs Randomized Withdrawal Period: Placebo; Test type: Superiority; p = 0.0022, Cochran-Mantel-Haenszel — 95% CI and p-value were analyzed using a Cochran-Mantel-Haenszel test adjusted by oral corticosteroid use and diagnosis of recurrent idiopathic pericarditis at run-in baseline; Odds Ratio (OR) = 8.370, 95% CI 2-sided [1.317 to 53.188]

6. Secondary Outcome: Percentage of Participants Who Maintained Clinical Response at Week 8 of the RW Period
Description: Participants were asked to select the score that best describes their average level of pericarditis pain over the previous 24 hours using an 11-point numerical rating scale (NRS), where zero (0) indicates 'no pain' and ten (10) indicates 'pain as bad as it could be'. Clinical response was defined as a weekly average of daily pericarditis pain on the NRS ≤ 2.0 and C-reactive protein (CRP) level ≤ 0.5 mg/dL, and on monotherapy of randomized study drug at Week 8.
Time Frame: RW Period Week 8
Population: ITT Week 8 Analysis Set: All participants randomized at least 8 weeks before data cutoff.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomized Withdrawal Period: Rilonacept | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 27 | 31
percentage of participants | 77.8 [57.7 to 91.4] | 25.8 [11.9 to 44.6]
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: Rilonacept vs Randomized Withdrawal Period: Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 5, analysis 1]; Odds Ratio (OR) = 10.906, 95% CI 2-sided [3.051 to 38.981]

7. Secondary Outcome: Percentage of Days With No or Minimal Pericarditis Pain at Week 24 of the RW Period
Description: Participants were asked to select the score that best describes their average level of pericarditis pain over the previous 24 hours using an 11-point numerical rating scale (NRS), where zero (0) indicates 'no pain' and ten (10) indicates 'pain as bad as it could be'. No or minimal pain was defined as non-missing NRS ≤ 2.
  The percentage of days with no or minimal pericarditis pain in the first 24 weeks was calculated for each participant using 24×7 as the denominator. Missing values in pain diary were counted as 0 day with no or minimal pain. Days of using oral rescue therapy or corticosteroid count as 0 day with no or minimal pain. If bailout rilonacept was used, each administration (loading dose or not) was counted as 7 days without qualifying no or minimal pain.
Time Frame: RW Period Week 24
Population: ITT Week 24 Analysis Set: All participants randomized at least 24 weeks before data cutoff.
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Randomized Withdrawal Period: Rilonacept | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 17 | 15
percentage of days | 100.6 (8.02) | 48.7 (7.64)
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: Rilonacept vs Randomized Withdrawal Period: Placebo; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS mean difference = 51.9, 95% CI 2-sided [33.8 to 70.1] — Least squares mean difference (rilonacept - placebo)

8. Secondary Outcome: Percentage of Days With No or Minimal Pericarditis Pain at Week 8 of the RW Period
Description: Participants were asked to select the score that best describes their average level of pericarditis pain over the previous 24 hours using an 11-point numerical rating scale (NRS), where zero (0) indicates 'no pain' and ten (10) indicates 'pain as bad as it could be'. No or minimal pain was defined as non-missing NRS ≤ 2.
  The percentage of days with no or minimal pericarditis pain in the first 24 weeks was calculated for each participant using 8×7 as the denominator. Missing values in pain diary were counted as 0 day with no or minimal pain. Days of using oral rescue therapy or corticosteroid count as 0 day with no or minimal pain. If bailout rilonacept was used, each administration (loading dose or not) was counted as 7 days without qualifying no or minimal pain.
Time Frame: RW Period Week 8
Population: ITT Week 8 Analysis Set: All participants randomized at least 8 weeks before data cutoff.
Measure: Least Squares Mean (Standard Error); unit: percentage of days
Arm/Group | Randomized Withdrawal Period: Rilonacept | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 27 | 31
percentage of days | 97.9 (7.64) | 57.3 (7.19)
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: Rilonacept vs Randomized Withdrawal Period: Placebo; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; LS mean difference = 40.5, 95% CI 2-sided [25.3 to 55.8] — Least squares mean difference (rilonacept - placebo)

9. Secondary Outcome: Percentage of Participants With Absent or Minimal Pericarditis Symptoms at Week 24 of the RW Period Based on the PGIPS
Description: Percentage of participants with no or minimal pericarditis symptoms at Week 24, based on the PGIPS, a single-item measure of the participant's impression of the overall severity of pericarditis symptoms at the time the questionnaire is administered using a 7-point rating scale ranging from absent (0=no recurrent pericarditis symptoms) to very severe (6=recurrent pericarditis symptoms cannot be ignored and markedly limits daily activities).
  The exact 95% CI is calculated with randomization strata pooled. Participants who had received bailout rilonacept or rescue medication before the time point were considered nonresponders.
Time Frame: RW Period Week 24
Population: ITT Week 24 Analysis Set: All participants randomized at least 24 weeks before data cutoff.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomized Withdrawal Period: Rilonacept | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 17 | 15
percentage of participants | 88.2 [63.6 to 98.5] | 20.0 [4.3 to 48.1]
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: Rilonacept vs Randomized Withdrawal Period: Placebo; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel — 95% CI and p-value are analyzed using a Cochran-Mantel-Haenszel (CMH) test adjusted by oral corticosteroid use at RI baseline; Odds Ratio (OR) = 30.522, 95% CI 2-sided [4.262 to 218.552]

10. Secondary Outcome: Percentage of Participants With Absent or Minimal Pericarditis Symptoms at Week 8 of the RW Period Based on the PGIPS
Description: Percentage of participants with no or minimal pericarditis symptoms at Week 16, based on the Patient Global Impression of Pericarditis Severity (PGI-PS). The PGI-PS is a single-item measure of the participant's impression of the overall severity of pericarditis symptoms at the time the questionnaire is administered, using a 7-point rating scale ranging from absent (no recurrent pericarditis symptoms) to very severe (recurrent pericarditis symptoms cannot be ignored).
  The exact 95% CI is calculated with randomization strata pooled. Participants who had received bailout rilonacept or rescue medication before the time point were considered nonresponders.
Time Frame: RW Period Week 8
Population: ITT Week 8 Analysis Set: All participants randomized at least 8 weeks before data cutoff.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomized Withdrawal Period: Rilonacept | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 27 | 31
percentage of participants | 85.2 [66.3 to 95.8] | 32.3 [16.7 to 51.4]
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: Rilonacept vs Randomized Withdrawal Period: Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Odds Ratio (OR) = 14.432, 95% CI 2-sided [3.439 to 60.574]

11. Secondary Outcome: Percentage of Participants Without Pericarditis Recurrence in the First 24 Weeks of the RW Period
Description: Pericarditis recurrence is defined as the recurrence of typical pericarditis pain associated with supportive objective evidence of pericarditis. At any time during the RW period, participants who experienced a suspected recurrence of pericarditis symptoms reported to the study site/clinic for a scheduled or unscheduled visit, during which clinical assessments were performed to gather all the necessary diagnostic data to confirm or rule out the presence of pericarditis recurrence. A pericarditis recurrence event adjudication package was then prepared for adjudication by CEC. Kaplan-Meier estimate.
Time Frame: up to 24 weeks in the RW Period
Population: ITT Analysis Set: all participants who were randomized in the RW period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomized Withdrawal Period: Rilonacept | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 30 | 31
percentage of participants | 95.7 [72.9 to 99.4] | 19.9 [6.5 to 38.6]
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: Rilonacept vs Randomized Withdrawal Period: Placebo; Test type: Superiority; p < 0.0001, normal approximation; Difference = 75.7, 95% CI 2-sided [56.8 to 94.6]

12. Secondary Outcome: Time to Pericarditis Pain ≥ 4 on the NRS in the RW Period
Description: Participants were asked to select the score that best described their average level of pericarditis pain over the previous 24 hours using an 11-point numerical rating scale (NRS), where zero (0) indicates 'no pain' and ten (10) indicates 'pain as bad as it could be'.
Time Frame: RW Period (mean 24.8 weeks)
Population: ITT Analysis Set: all participants who were randomized in the RW period.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Randomized Withdrawal Period: Rilonacept | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 30 | 31
weeks | NA [33.1 to NA] — Median not reached due to low events. | 4.1 [2.9 to 6.6]
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: Rilonacept vs Randomized Withdrawal Period: Placebo; Test type: Superiority; p < 0.0001, Log Rank — Two-sided p-value is from the log-rank test stratified by oral corticosteroid use at run-in baseline; Hazard Ratio (HR) = 0.13, 95% CI 2-sided [0.05 to 0.32] — Calculated based on a Cox proportional hazards model with treatment as covariate and stratified by oral corticosteroid use at run-in baseline

13. Secondary Outcome: Time to CRP Level ≥ 1 mg/dL in the RW Period
Description: Kaplan-Meier estimate.
Time Frame: RW Period (mean 24.8 weeks)
Population: ITT Analysis Set: all participants who were randomized in the RW period.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Randomized Withdrawal Period: Rilonacept | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 30 | 31
weeks | NA [NA to NA] — Median not reached due to low number of participants with CRP ≥ 1 mg/dL. | 6.9 [4.0 to 10.1]
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: Rilonacept vs Randomized Withdrawal Period: Placebo; Test type: Superiority; p < 0.0001, Log Rank — Two-sided p-value is from the log-rank test stratified by oral corticosteroid use at run-in baseline; Hazard Ratio (HR) = 0.07, 95% CI 2-sided [0.02 to 0.22] — [estimate comment as in outcome 12, analysis 1]

14. Secondary Outcome: Time to Pericardial Rub in the RW Period
Description: Kaplan-Meier estimate. A pericardial rub (also called a pericardial friction rub) is an audible medical sign used in the diagnosis of pericarditis.
Time Frame: RW Period (mean 24.8 weeks)
Population: ITT Analysis Set: all participants who were randomized in the RW period.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Randomized Withdrawal Period: Rilonacept | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 30 | 31
weeks | NA [NA to NA] — Not estimable due to low number of participants with an event. | NA [NA to NA] — Not estimable due to low number of participants with an event.
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: Rilonacept vs Randomized Withdrawal Period: Placebo; Test type: Superiority; p = 0.7447, Log Rank — Two-sided p-value is from the log-rank test without stratification by randomization strata; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.12 to 4.46] — Calculated based on a Cox proportional-hazards model with treatment as covariate and without stratification by randomization strata

15. Secondary Outcome: Time to Widespread ST-segment Elevation or PR-segment Depression on Electrocardiogram (ECG) in the RW Period
Description: Kaplan-Meier estimate. ST-segment elevation and PR-segment depression are ECG changes in the evolution of acute pericarditis.
Time Frame: RW Period (mean 24.8 weeks)
Population: ITT Analysis Set: all participants who were randomized in the RW period.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Randomized Withdrawal Period: Rilonacept | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 30 | 31
weeks | NA [NA to NA] — Not estimable due to low number of participants with an event. | NA [NA to NA] — Not estimable due to low number of participants with an event.
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: Rilonacept vs Randomized Withdrawal Period: Placebo; Test type: Superiority; p = 0.2066, Log Rank — Two-sided p-value is from the log-rank test without stratification by randomization strata; Hazard Ratio (HR) = 0.36, 95% CI 2-sided [0.07 to 1.87] — [estimate comment as in outcome 14, analysis 1]

16. Secondary Outcome: Time to New or Worsening Pericardial Effusion on Echocardiography (ECHO) in the RW Period
Description: Pericardial effusion based on ECHO was evaluated by the central laboratory during the RW period. Kaplan-Meier estimate.
Time Frame: RW Period (mean 24.8 weeks)
Population: ITT Analysis Set: all participants who were randomized in the RW period.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Randomized Withdrawal Period: Rilonacept | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 30 | 31
weeks | NA [NA to NA] — Not estimable due to low number of participants with an event. | NA [NA to NA] — Not estimable due to low number of participants with an event.
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: Rilonacept vs Randomized Withdrawal Period: Placebo; Test type: Superiority; p = 0.0059, Log Rank — Two-sided p-value is from the log-rank test without stratification by randomization strata; Hazard Ratio (HR) = 0.00, 95% CI 2-sided [lower limit 0.00] (Not estimable due to low number of participants with an event.)

17. Secondary Outcome: Number of Participants in ECHO Pericardial Effusion Size Categories at RW Period Baseline, RW Week 24 and Worst Post-baseline in the RW Period
Description: Pericardial effusion based on ECHO was evaluated by the central laboratory during the RW period. "None or trivial/physiologic" is considered to be normal. The "RW Worst Post-baseline" category denotes the largest size of pericardial effusion category in which a participant was reported at any time during the RW period (post-baseline).
Time Frame: RW Period Baseline, RW Period Week 24, RW Period (mean 24.8 weeks)
Population: ITT Analysis Set: all participants who were randomized in the RW period. Participants with a non-missing value at given time point.
Measure: Count of Participants; unit: Participants
Groups:
- Randomized Withdrawal Period: Rilonacept, Before Bailout Rilonacept: Double-blind rilonacept 160 mg (or 2.2 mg/kg in pediatric participants ≥ 12 and < 18 years old) SC injections once weekly.
- Randomized Withdrawal Period: Rilonacept, Including Bailout Rilonacept: Double-blind rilonacept 160 mg (or 2.2 mg/kg in pediatric participants ≥ 12 and < 18 years old) SC injections once weekly.
  Participants with pericarditis recurrence who meet the protocol criteria for bailout rilonacept (report at least 1 day with pericarditis pain ≥4 on the 11-point NRS and have 1 CRP value ≥ 1 mg/dL [either on the same day or separated by no more than 7 days]) receive bailout rilonacept (2 open-label injections of 160 mg rilonacept [or 4.4 mg/kg for pediatric participants]) irrespective of randomized treatment assignment and as soon as at least 5 days have passed since the last study drug injection.
- Randomized Withdrawal Period: Placebo, Before Bailout Rilonacept: Double-blind placebo SC injections once weekly.
- Randomized Withdrawal Period: Placebo, Including Bailout Rilonacept: Double-blind placebo SC injections once weekly.
  Participants with pericarditis recurrence who meet the protocol criteria for bailout rilonacept (report at least 1 day with pericarditis pain ≥4 on the 11-point NRS and have 1 CRP value ≥ 1 mg/dL [either on the same day or separated by no more than 7 days]) receive bailout rilonacept (2 open-label injections of 160 mg rilonacept [or 4.4 mg/kg for pediatric participants]) irrespective of randomized treatment assignment and as soon as at least 5 days have passed since the last study drug injection.
Arm/Group | Randomized Withdrawal Period: Rilonacept, Before Bailout Rilonacept | Randomized Withdrawal Period: Rilonacept, Including Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Before Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Including Bailout Rilonacept
Number analyzed (Participants) | 30 | 30 | 31 | 31
Participants
  RW Baseline: None or Trivial/Physiologic | 28 | 28 | 30 | 30
  RW Baseline: Small | 1 | 1 | 1 | 1
  RW Baseline: Moderate | 1 | 1 | 0 | 0
  RW Baseline: Large | 0 | 0 | 0 | 0
  RW Baseline: Very Large | 0 | 0 | 0 | 0
  RW Baseline: Missing/Not Done | 0 | 0 | 0 | 0
  RW Week 24: number analyzed (Participants) | 12 | 12 | 3 | 13
  RW Week 24: None or Trivial/Physiologic | 12 | 12 | 3 | 13
  RW Week 24: Small | 0 | 0 | 0 | 0
  RW Week 24: Moderate | 0 | 0 | 0 | 0
  RW Week 24: Large | 0 | 0 | 0 | 0
  RW Week 24: Very Large | 0 | 0 | 0 | 0
  RW Week 24: Missing/Not Done | 0 | 0 | 0 | 0
  RW Worst Post-baseline: number analyzed (Participants) | 28 | 28 | 19 | 28
  RW Worst Post-baseline: None or Trivial/Physiologic | 28 | 28 | 14 | 20
  RW Worst Post-baseline: Small | 0 | 0 | 4 | 7
  RW Worst Post-baseline: Moderate | 0 | 0 | 1 | 1
  RW Worst Post-baseline: Large | 0 | 0 | 0 | 0
  RW Worst Post-baseline: Very Large | 0 | 0 | 0 | 0
  RW Worst Post-baseline: Missing/Not Done | 0 | 0 | 0 | 0

18. Secondary Outcome: Change From RW Period Baseline Over Time in CRP Levels in RW Period
Description: Estimated from ANCOVA models including treatment arm as fix effect, baseline value, baseline value by treatment interaction, randomization strata as covariates.
Time Frame: RW Period Baseline, RW Period Weeks 4, 8, 12, 16, 20, 24, 32, 40, 48, 56
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Randomized Withdrawal Period: Rilonacept, Before Bailout Rilonacept | Randomized Withdrawal Period: Rilonacept, Including Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Before Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Including Bailout Rilonacept
Number analyzed (Participants) | 30 | 30 | 31 | 31
mg/dL
  Change at RW Week 4: number analyzed (Participants) | 27 | 27 | 20 | 29
  Change at RW Week 4 | -0.01 (0.058) | -0.05 (1.112) | 0.15 (0.061) | 1.46 (0.861)
  Change at RW Week 8: number analyzed (Participants) | 22 | 22 | 14 | 26
  Change at RW Week 8 | 0.12 (0.308) | 0.11 (0.300) | 0.45 (0.331) | 0.25 (0.246)
  Change at RW Week 12: number analyzed (Participants) | 20 | 20 | 7 | 21
  Change at RW Week 12 | 0.04 (0.034) | -0.04 (0.085) | 0.03 (0.043) | 0.08 (0.077)
  Change at RW Week 16: number analyzed (Participants) | 21 | 21 | 5 | 20
  Change at RW Week 16 | 0.40 (0.148) | 0.27 (0.119) | 0.04 (0.227) | 0.18 (0.109)
  Change at RW Week 20: number analyzed (Participants) | 16 | 16 | 3 | 14
  Change at RW Week 20 | -0.04 (0.048) | -0.10 (0.181) | 0.10 (0.083) | 0.16 (0.174)
  Change at RW Week 24: number analyzed (Participants) | 15 | 15 | 3 | 14
  Change at RW Week 24 | -0.04 (0.032) | -0.05 (0.047) | 0.06 (0.056) | 0.02 (0.045)
  Change at RW Week 32: number analyzed (Participants) | 11 | 12 | 1 | 11
  Change at RW Week 32 | -0.05 (0.016) | -0.02 (0.059) | NA (NA) — Not estimable due to statistical analysis system (SAS) algorithms. | 0.07 (0.055)
  Change at RW Week 40: number analyzed (Participants) | 5 | 6 | 1 | 6
  Change at RW Week 40 | 0.04 (0.010) | 0.08 (0.298) | NA (NA) — Not estimable due to SAS algorithms. | 0.74 (0.290)
  Change at RW Week 48: number analyzed (Participants) | 4 | 5 | 0 | 2
  Change at RW Week 48 | 0.02 (0.000) | -0.03 (0.008) |  | 0.06 (0.017)
  Change at RW Week 56: number analyzed (Participants) | 0 | 0 | 0 | 1
  Change at RW Week 56 |  |  |  | 0.00 (NA) — 1 participant in arm at time point

19. Secondary Outcome: Change From RW Period Baseline Over Time in Weekly Average of Pericarditis Pain in the RW Period
Description: Participants were asked to select the score that best described their average level of pericarditis pain over the previous 24 hours using an 11-point numerical rating scale (NRS), where zero (0) indicates 'no pain' and ten (10) indicates 'pain as bad as it could be'. Estimated from ANCOVA models including treatment arm as fix effect, baseline value, baseline value by treatment interaction, randomization strata as covariates.
Time Frame: RW Period Baseline, RW Period Weeks 1-50, 54
Population: as for outcome 17
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Randomized Withdrawal Period: Rilonacept, Before Bailout Rilonacept | Randomized Withdrawal Period: Rilonacept, Including Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Before Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Including Bailout Rilonacept
Number analyzed (Participants) | 30 | 30 | 31 | 31
units on a scale
  Change at RW Week 1: number analyzed (Participants) | 29 | 29 | 31 | 31
  Change at RW Week 1 | -0.08 (0.103) | -0.08 (0.103) | 0.17 (0.099) | 0.17 (0.099)
  Change at RW Week 2: number analyzed (Participants) | 29 | 29 | 29 | 31
  Change at RW Week 2 | -0.21 (0.237) | -0.25 (0.273) | 0.57 (0.231) | 0.68 (0.263)
  Change at RW Week 3: number analyzed (Participants) | 27 | 27 | 27 | 31
  Change at RW Week 3 | -0.08 (0.296) | -0.15 (0.330) | 1.12 (0.278) | 1.29 (0.302)
  Change at RW Week 4: number analyzed (Participants) | 27 | 27 | 20 | 30
  Change at RW Week 4 | -0.16 (0.322) | -0.11 (0.468) | 1.05 (0.333) | 1.84 (0.428)
  Change at RW Week 5: number analyzed (Participants) | 26 | 26 | 17 | 29
  Change at RW Week 5 | -0.16 (0.314) | -0.21 (0.351) | 1.27 (0.332) | 1.34 (0.320)
  Change at RW Week 6: number analyzed (Participants) | 24 | 24 | 14 | 27
  Change at RW Week 6 | 0.22 (0.296) | 0.02 (0.310) | 0.96 (0.290) | 0.84 (0.265)
  Change at RW Week 7: number analyzed (Participants) | 25 | 25 | 14 | 29
  Change at RW Week 7 | 0.06 (0.273) | 0.12 (0.248) | 0.87 (0.304) | 0.86 (0.224)
  Change at RW Week 8: number analyzed (Participants) | 25 | 25 | 13 | 26
  Change at RW Week 8 | 0.10 (0.226) | 0.11 (0.205) | 0.77 (0.253) | 0.58 (0.189)
  Change at RW Week 9: number analyzed (Participants) | 25 | 25 | 9 | 23
  Change at RW Week 9 | -0.24 (0.310) | 0.05 (0.320) | 1.45 (0.402) | 1.10 (0.301)
  Change at RW Week 10: number analyzed (Participants) | 23 | 23 | 9 | 24
  Change at RW Week 10 | -0.17 (0.270) | -0.21 (0.262) | 1.11 (0.343) | 0.62 (0.240)
  Change at RW Week 11: number analyzed (Participants) | 23 | 23 | 9 | 23
  Change at RW Week 11 | -0.20 (0.200) | -0.16 (0.272) | 0.43 (0.267) | 0.46 (0.250)
  Change at RW Week 12: number analyzed (Participants) | 22 | 22 | 8 | 24
  Change at RW Week 12 | 0.07 (0.174) | -0.03 (0.248) | 0.36 (0.235) | 0.32 (0.225)
  Change at RW Week 13: number analyzed (Participants) | 22 | 22 | 7 | 23
  Change at RW Week 13 | -0.02 (0.331) | 0.06 (0.256) | 0.25 (0.386) | 0.07 (0.220)
  Change at RW Week 14: number analyzed (Participants) | 22 | 22 | 7 | 22
  Change at RW Week 14 | 0.14 (0.186) | 0.08 (0.185) | 0.24 (0.262) | 0.06 (0.170)
  Change at RW Week 15: number analyzed (Participants) | 21 | 21 | 6 | 22
  Change at RW Week 15 | 0.32 (0.109) | 0.19 (0.149) | -0.08 (0.235) | 0.15 (0.136)
  Change at RW Week 16: number analyzed (Participants) | 19 | 19 | 5 | 18
  Change at RW Week 16 | 0.12 (0.110) | -0.07 (0.167) | NA (NA) — Not estimable due to SAS algorithms. | 0.09 (0.153)
  Change at RW Week 17: number analyzed (Participants) | 17 | 17 | 5 | 18
  Change at RW Week 17 | 0.19 (0.129) | 0.01 (0.183) | NA (NA) — Not estimable due to SAS algorithms. | 0.05 (0.165)
  Change at RW Week 18: number analyzed (Participants) | 15 | 15 | 5 | 16
  Change at RW Week 18 | 0.13 (0.149) | 0.05 (0.157) | NA (NA) — Not estimable due to SAS algorithms. | -0.05 (0.131)
  Change at RW Week 19: number analyzed (Participants) | 16 | 16 | 5 | 17
  Change at RW Week 19 | 0.04 (0.149) | -0.05 (0.167) | NA (NA) — Not estimable due to SAS algorithms. | -0.04 (0.139)
  Change at RW Week 20: number analyzed (Participants) | 17 | 17 | 3 | 14
  Change at RW Week 20 | -0.08 (0.111) | -0.22 (0.228) | NA (NA) — Not estimable due to SAS algorithms. | 0.30 (0.226)
  Change at RW Week 21: number analyzed (Participants) | 17 | 17 | 3 | 14
  Change at RW Week 21 | 0.04 (0.156) | 0.02 (0.162) | NA (NA) — Not estimable due to SAS algorithms. | 0.23 (0.160)
  Change at RW Week 22: number analyzed (Participants) | 16 | 16 | 3 | 14
  Change at RW Week 22 | -0.08 (0.097) | -0.12 (0.124) | NA (NA) — Not estimable due to SAS algorithms. | 0.01 (0.120)
  Change at RW Week 23: number analyzed (Participants) | 15 | 15 | 3 | 14
  Change at RW Week 23 | -0.01 (0.103) | -0.03 (0.145) | NA (NA) — Not estimable due to SAS algorithms. | -0.01 (0.140)
  Change at RW Week 24: number analyzed (Participants) | 15 | 15 | 3 | 14
  Change at RW Week 24 | 0.02 (0.122) | -0.04 (0.138) | NA (NA) — Not estimable due to SAS algorithms. | 0.02 (0.132)
  Change at RW Week 25: number analyzed (Participants) | 14 | 14 | 3 | 12
  Change at RW Week 25 | 0.12 (0.122) | 0.09 (0.109) | NA (NA) — Not estimable due to SAS algorithms. | 0.13 (0.110)
  Change at RW Week 26: number analyzed (Participants) | 15 | 15 | 3 | 11
  Change at RW Week 26 | 0.19 (0.145) | 0.16 (0.127) | NA (NA) — Not estimable due to SAS algorithms. | 0.29 (0.131)
  Change at RW Week 27: number analyzed (Participants) | 15 | 15 | 3 | 12
  Change at RW Week 27 | 0.23 (0.193) | 0.16 (0.154) | NA (NA) — Not estimable due to SAS algorithms. | 0.15 (0.157)
  Change at RW Week 28: number analyzed (Participants) | 14 | 14 | 3 | 12
  Change at RW Week 28 | 0.38 (0.449) | 0.33 (0.339) | NA (NA) — Not estimable due to SAS algorithms. | 0.18 (0.340)
  Change at RW Week 29: number analyzed (Participants) | 12 | 13 | 2 | 11
  Change at RW Week 29 | 0.26 (0.160) | 0.29 (0.233) | NA (NA) — Not estimable due to SAS algorithms. | 0.12 (0.227)
  Change at RW Week 30: number analyzed (Participants) | 11 | 12 | 2 | 11
  Change at RW Week 30 | 0.25 (0.296) | 0.39 (0.259) | NA (NA) — Not estimable due to SAS algorithms. | 0.64 (0.250)
  Change at RW Week 31: number analyzed (Participants) | 11 | 12 | 2 | 11
  Change at RW Week 31 | 0.06 (0.110) | 0.02 (0.109) | NA (NA) — Not estimable due to SAS algorithms. | 0.33 (0.105)
  Change at RW Week 32: number analyzed (Participants) | 9 | 10 | 2 | 11
  Change at RW Week 32 | 0.47 (0.081) | 0.20 (0.141) | NA (NA) — Not estimable due to SAS algorithms. | 0.23 (0.118)
  Change at RW Week 33: number analyzed (Participants) | 8 | 9 | 1 | 10
  Change at RW Week 33 | 0.62 (0.016) | 0.31 (0.167) | NA (NA) — Not estimable due to SAS algorithms. | 0.20 (0.151)
  Change at RW Week 34: number analyzed (Participants) | 6 | 7 | 1 | 9
  Change at RW Week 34 | 1.64 (0.086) | 0.95 (0.387) | NA (NA) — Not estimable due to SAS algorithms. | 0.27 (0.329)
  Change at RW Week 35: number analyzed (Participants) | 6 | 7 | 1 | 9
  Change at RW Week 35 | 0.75 (0.055) | 0.62 (0.347) | NA (NA) — Not estimable due to SAS algorithms. | 0.11 (0.295)
  Change at RW Week 36: number analyzed (Participants) | 7 | 8 | 1 | 8
  Change at RW Week 36 | 0.25 (0.093) | 0.15 (0.348) | NA (NA) — Not estimable due to SAS algorithms. | 0.20 (0.346)
  Change at RW Week 37: number analyzed (Participants) | 6 | 7 | 1 | 7
  Change at RW Week 37 | -0.02 (0.243) | -0.13 (0.404) | NA (NA) — Not estimable due to SAS algorithms. | 0.16 (0.367)
  Change at RW Week 38: number analyzed (Participants) | 6 | 7 | 1 | 7
  Change at RW Week 38 | 0.56 (0.022) | 0.40 (0.177) | NA (NA) — Not estimable due to SAS algorithms. | 0.04 (0.162)
  Change at RW Week 39: number analyzed (Participants) | 5 | 6 | 1 | 6
  Change at RW Week 39 | 0.96 (0.260) | 0.55 (0.578) | NA (NA) — Not estimable due to SAS algorithms. | 0.51 (0.592)
  Change at RW Week 40: number analyzed (Participants) | 4 | 5 | 1 | 6
  Change at RW Week 40 | NA (NA) — Not estimable due to SAS algorithms. | 0.17 (1.253) | NA (NA) — Not estimable due to SAS algorithms. | 0.44 (1.002)
  Change at RW Week 41: number analyzed (Participants) | 5 | 6 | 0 | 5
  Change at RW Week 41 | 0.92 (0.293) | 0.72 (0.723) |  | 0.91 (0.939)
  Change at RW Week 42: number analyzed (Participants) | 5 | 6 | 0 | 4
  Change at RW Week 42 | 0.77 (0.488) | 0.79 (0.262) |  | 0.60 (0.342)
  Change at RW Week 43: number analyzed (Participants) | 5 | 6 | 0 | 4
  Change at RW Week 43 | 1.03 (0.619) | 0.87 (0.449) |  | 0.88 (0.587)
  Change at RW Week 44: number analyzed (Participants) | 5 | 6 | 0 | 5
  Change at RW Week 44 | 0.84 (0.553) | 0.64 (0.590) |  | 0.75 (0.766)
  Change at RW Week 45: number analyzed (Participants) | 5 | 6 | 0 | 2
  Change at RW Week 45 | 0.77 (0.567) | 0.85 (0.384) |  | 3.77 (1.564)
  Change at RW Week 46: number analyzed (Participants) | 4 | 5 | 0 | 1
  Change at RW Week 46 | 0.18 (0.680) | 0.39 (0.471) |  | NA (NA) — Not estimable due to SAS algorithms.
  Change at RW Week 47: number analyzed (Participants) | 4 | 5 | 0 | 2
  Change at RW Week 47 | 0.07 (0.000) | 0.16 (0.261) |  | 3.10 (1.070)
  Change at RW Week 48: number analyzed (Participants) | 3 | 4 | 0 | 2
  Change at RW Week 48 | 0.03 (0.000) | 0.32 (0.273) |  | 6.18 (1.490)
  Change at RW Week 49: number analyzed (Participants) | 2 | 3 | 0 | 2
  Change at RW Week 49 | -0.50 (0.000) | -0.13 (0.115) |  | 5.77 (0.630)
  Change at RW Week 50: number analyzed (Participants) | 1 | 1 | 0 | 0
  Change at RW Week 50 | 0.00 (NA) — 1 participant | 0.00 (NA) — 1 participant |  |
  Change at RW Week 54: number analyzed (Participants) | 0 | 0 | 0 | 1
  Change at RW Week 54 |  |  |  | 0.58 (0.000)

20. Secondary Outcome: Percentage of Participants With Absent or Minimal Pericarditis Symptoms Over Time After RW Period Week 24 Based on the PGIPS
Description: The PGIPS, a single-item measure of the participant's impression of the overall severity of pericarditis symptoms at the time the questionnaire is administered using a 7-point rating scale ranging from absent (0=no recurrent pericarditis symptoms) to very severe (6=recurrent pericarditis symptoms cannot be ignored and markedly limits daily activities).
  The exact 95% CI is calculated with randomization strata pooled. Participants who had received bailout rilonacept or rescue medication before the time point were considered nonresponders.
Time Frame: RW Period Weeks 32, 40, 48, 56
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomized Withdrawal Period: Rilonacept, Before Bailout Rilonacept | Randomized Withdrawal Period: Rilonacept, Including Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Before Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Including Bailout Rilonacept
Number analyzed (Participants) | 11 | 12 | 2 | 10
percentage of participants
  Week 32 | 90.9 [58.72 to 99.77] | 83.3 [51.59 to 97.91] | 50.0 [1.26 to 98.74] | 70.0 [34.75 to 93.33]
  Week 40: number analyzed (Participants) | 5 | 6 | 1 | 6
  Week 40 | 60.0 [14.66 to 94.73] | 66.7 [22.28 to 95.67] | 100 [2.50 to 100.00] | 83.3 [35.88 to 99.58]
  Week 48: number analyzed (Participants) | 2 | 2 | 0 | 2
  Week 48 | 100 [15.81 to 100.00] | 100 [15.81 to 100.00] |  | 50.0 [1.26 to 98.74]
  Week 56: number analyzed (Participants) | 0 | 0 | 0 | 1
  Week 56 |  |  |  | 100 [2.50 to 100.00]

21. Secondary Outcome: Percentage of Participants With Absent or Minimal Pericarditis Activity Over Time in the RW Period Based on the Physician Global Assessment of Pericarditis Activity (PGA-PA)
Description: The PGA-PA is a single-item, clinician-reported outcome measure that Investigators use to rate their impression of the patient's overall pericarditis disease activity at the time the assessment is completed, using a rating scale ranging from absent to very severe. The Investigator selected the box that best described a participant's pericarditis activity at the time of occurrence of the assessment: Absent, Minimal, Mild, Moderate, Moderately Severe, Severe, Very Severe.
Time Frame: RW Period Baseline, RW Period Weeks 8, 16, 24, 32, 40, 48, 56
Population: as for outcome 17
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomized Withdrawal Period: Rilonacept, Before Bailout Rilonacept | Randomized Withdrawal Period: Rilonacept, Including Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Before Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Including Bailout Rilonacept
Number analyzed (Participants) | 30 | 30 | 31 | 31
percentage of participants
  Baseline | 96.7 [82.78 to 99.92] | 96.7 [82.78 to 99.92] | 100 [88.78 to 100.00] | 100 [88.78 to 100.00]
  Week 8: number analyzed (Participants) | 23 | 23 | 14 | 27
  Week 8 | 100 [85.18 to 100.00] | 100 [85.18 to 100.00] | 71.4 [41.90 to 91.61] | 85.2 [66.27 to 95.81]
  Week 16: number analyzed (Participants) | 20 | 20 | 5 | 20
  Week 16 | 95.0 [75.13 to 99.87] | 95.0 [75.13 to 99.87] | 100 [47.82 to 100.00] | 95.0 [75.13 to 99.87]
  Week 24: number analyzed (Participants) | 15 | 15 | 3 | 14
  Week 24 | 100 [78.20 to 100.00] | 100 [78.20 to 100.00] | 100 [29.24 to 100.00] | 100 [76.84 to 100.00]
  Week 32: number analyzed (Participants) | 11 | 12 | 2 | 11
  Week 32 | 90.9 [58.72 to 99.77] | 83.3 [51.59 to 97.91] | 50.0 [1.26 to 98.74] | 90.9 [58.72 to 99.77]
  Week 40: number analyzed (Participants) | 3 | 4 | 1 | 6
  Week 40 | 66.7 [9.43 to 99.16] | 75.0 [19.41 to 99.37] | 100 [2.50 to 100.00] | 100 [54.07 to 100.00]
  Week 48: number analyzed (Participants) | 2 | 2 | 0 | 2
  Week 48 | 50.0 [1.26 to 98.74] | 50.0 [1.26 to 98.74] |  | 50.0 [1.26 to 98.74]
  Week 56: number analyzed (Participants) | 0 | 0 | 0 | 1
  Week 56 |  |  |  | 100 [2.50 to 100.00]

22. Secondary Outcome: Change From RW Period Baseline in Short Form-36 (SF-36) Physical and Mental Component Scores at RW Period Week 24
Description: The SF-36 determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 primarily contribute to the physical component summary (PCS) score of the SF-36. Items 5-8 primarily contribute to the mental component summary (MCS) score of the SF-36. Scores on each item are summed and averaged (range: 0=worst to 100=best) with higher scores indicating better health. Increases from baseline indicate improvement.
Time Frame: RW Period Baseline, RW Period Week 24
Population: ITT Analysis Set: all participants who were randomized in the RW period. Participants 18 years and older with a non-missing value at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Withdrawal Period: Rilonacept, Before Bailout Rilonacept | Randomized Withdrawal Period: Rilonacept, Including Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Before Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Including Bailout Rilonacept
Number analyzed (Participants) | 15 | 15 | 3 | 14
score on a scale
  Change at RW Week 24 in PCS | 0.427 (5.8566) | 0.427 (5.8566) | 0.363 (2.3866) | 0.354 (2.7169)
  Change at RW Week 24 in MCS | 3.081 (11.3204) | 3.081 (11.3204) | -0.050 (2.7318) | -0.575 (5.5922)

23. Secondary Outcome: Change From RW Baseline in SF-36 Individual Scores at RW Period Week 24
Description: The SF-36 determines participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Scores on each item are summed and averaged (range: 0=worst to 100=best) with higher scores indicating better health. Increases from baseline indicate improvement.
Time Frame: RW Period Baseline, RW Period Week 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Withdrawal Period: Rilonacept, Before Bailout Rilonacept | Randomized Withdrawal Period: Rilonacept, Including Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Before Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Including Bailout Rilonacept
Number analyzed (Participants) | 15 | 15 | 3 | 14
score on a scale
  Change at RW Week 24 in Physical Functioning | 2.427 (5.3887) | 2.427 (5.3887) | -0.637 (1.1027) | 0.273 (4.0332)
  Change at RW Week 24 in Role Physical | 2.995 (5.7997) | 2.995 (5.7997) | 1.500 (2.5981) | 1.123 (3.4967)
  Change at RW Week 24 in Bodily Pain | -0.485 (9.7799) | -0.485 (9.7799) | 0.807 (5.2864) | 0.921 (6.2063)
  Change at RW Week 24 in General Health | -0.919 (4.9051) | -0.919 (4.9051) | -1.587 (5.9895) | -1.901 (6.8070)
  Change at RW Week 24 in Vitality | 3.168 (9.8845) | 3.168 (9.8845) | 1.980 (6.8589) | 0.636 (6.1850)
  Change at RW Week 24 in Social Functioning | 0.669 (8.6544) | 0.669 (8.6544) | 0.000 (0.0000) | -1.791 (4.2209)
  Change at RW Week 24 in Role Emotional | 3.251 (10.7297) | 3.251 (10.7297) | 0.000 (0.0000) | 0.249 (7.0264)
  Change at RW Week 24 in Mental Health | 3.314 (8.5900) | 3.314 (8.5900) | -0.873 (3.9923) | -0.187 (6.7646)

24. Secondary Outcome: Change From RW Period Baseline in the Short Form Health Survey-6 Domains (SF-6D) Utility Index Score at RW Period Week 24
Description: The SF-6D is calculated based on responses to 11 items on the SF-36, that correspond to 6 domains: physical functioning, role participation (combined role-physical and role-emotional), social functioning, bodily pain, mental health, and vitality. Individual respondents can be classified on any of 4 to 6 levels of functioning or limitations for each of 6 domains, thus allowing a respondent to be classified into any of 18,000 possible unique health states. Using a standard gamble technique, each of these health states were mapped onto the SF-6D index score, which ranges from 0.00 (worst possible health state/death) to 1.00 (best possible health state/perfect health).
Time Frame: RW Period Baseline, RW Period Week 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Withdrawal Period: Rilonacept, Before Bailout Rilonacept | Randomized Withdrawal Period: Rilonacept, Including Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Before Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Including Bailout Rilonacept
Number analyzed (Participants) | 15 | 15 | 3 | 14
score on a scale | 0.0385 (0.10879) | 0.0385 (0.10879) | -0.0027 (0.05705) | -0.0005 (0.09871)

25. Secondary Outcome: Change From RW Period Baseline in 5-level EuroQoL-5 Dimensions (EQ-5D-5L) Individual Scores and Index Value to RW Period Week 24
Description: The EQ-5D-5L is a self-reported health status questionnaire that consists of 6 questions used to calculate a health utility score for use in health economic analysis. There are 2 components to the EQ-5D-5L: a 5-item health state profile that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression used to obtain an Index Utility Score, as well as a visual analogue scale (VAS) that measures health state. Individual and index scores range from 0 to 1, with low scores representing a higher level of dysfunction. The VAS is designed to rate the participant's current health state on a scale from 0 to 100, where 0 represents the worst imaginable health state and 100 represents the best imaginable health state.
Time Frame: RW Period Baseline, RW Period Week 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Withdrawal Period: Rilonacept, Before Bailout Rilonacept | Randomized Withdrawal Period: Rilonacept, Including Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Before Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Including Bailout Rilonacept
Number analyzed (Participants) | 15 | 15 | 3 | 14
score on a scale
  Change at RW Week 24 in Mobility | -0.1 (0.52) | -0.1 (0.52) | 0.0 (0.00) | -0.1 (0.53)
  Change at RW Week 24 in Self-Care | -0.1 (0.26) | -0.1 (0.26) | 0.0 (0.00) | 0.1 (0.27)
  Change at RW Week 24 in Usual Activities | -0.1 (0.70) | -0.1 (0.70) | 0.0 (0.00) | 0.1 (0.36)
  Change at RW Week 24 in Pain/Discomfort | 0.1 (0.92) | 0.1 (0.92) | 0.0 (1.00) | 0.1 (0.47)
  Change at RW Week 24 in Anxiety/Depression | -0.1 (0.83) | -0.1 (0.83) | -0.3 (0.58) | 0.0 (0.55)
  Change at RW Week 24 in Index Score | 0.0033 (0.09812) | 0.0033 (0.09812) | 0.0413 (0.15635) | 0.0029 (0.08592)
  Change at RW Week 24 in VAS Score | 7.5 (17.32) | 7.5 (17.32) | 10.0 (10.15) | -8.3 (29.07)

26. Secondary Outcome: Change From RW Period Baseline in Insomnia Severity Index (ISI) Total Score at RW Period Week 24
Description: Participant's sleep quality was assessed with the ISI survey questionnaire. The ISI is a 7-item survey, with each question having 5 possible answers (none, mild, moderate, severe, or very severe), scored as 0, 1, 2, 3, or 4, respectively. Scores are summed for a total score, which ranges from 0 to 28. Lower scores are considered good, better, or healthy, and increasingly higher scores are considered to indicate greater insomnia.
  Clinical interpretation of the total score is as follows:
  0 to 7 = no clinically significant insomnia; 8 to 14 = subthreshold insomnia; 15 to 21 = clinical insomnia (moderate severity); 22 to 28 = clinical insomnia (severe).
Time Frame: RW Period Baseline, RW Period Week 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Withdrawal Period: Rilonacept, Before Bailout Rilonacept | Randomized Withdrawal Period: Rilonacept, Including Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Before Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Including Bailout Rilonacept
Number analyzed (Participants) | 15 | 15 | 3 | 14
score on a scale | -0.7 (4.75) | -0.7 (4.75) | -0.3 (3.79) | -0.2 (2.99)

27. Secondary Outcome: Change in ISI Categories From RW Period Baseline to RW Period Week 24
Description: as for outcome 26
Time Frame: RW Period Baseline (BL), RW Period Week (Wk) 24
Population: ITT Week 24 Analysis Set: All participants randomized at least 24 weeks before data cutoff. Participants 18 years or older
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Withdrawal Period: Rilonacept, Before Bailout Rilonacept | Randomized Withdrawal Period: Rilonacept, Including Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Before Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Including Bailout Rilonacept
Number analyzed (Participants) | 17 | 17 | 15 | 15
Participants
  BL No Clinically Significant Insomnia: number analyzed (Participants) | 12 | 12 | 11 | 11
  BL No Clinically Significant Insomnia: Wk 24 No Clinically Significant Insomnia | 7 | 7 | 2 | 9
  BL No Clinically Significant Insomnia: Wk 24 Subthreshold Insomnia | 3 | 3 | 1 | 1
  BL No Clinically Significant Insomnia: Wk 24 Clinical Insomnia, Moderate Severity | 0 | 0 | 0 | 0
  BL No Clinically Significant Insomnia: Wk 24 Clinical Insomnia, Severe | 0 | 0 | 0 | 0
  BL No Clinically Significant Insomnia: Wk 24 Missing | 2 | 2 | 8 | 1
  BL Subthreshold Insomnia: number analyzed (Participants) | 3 | 3 | 4 | 4
  BL Subthreshold Insomnia: Wk 24 No Clinically Significant Insomnia | 2 | 2 | 0 | 2
  BL Subthreshold Insomnia: Wk 24 Subthreshold Insomnia | 1 | 1 | 0 | 2
  BL Subthreshold Insomnia: Wk 24 Clinical Insomnia, Moderate Severity | 0 | 0 | 0 | 0
  BL Subthreshold Insomnia: Wk 24 Clinical Insomnia, Severe | 0 | 0 | 0 | 0
  BL Subthreshold Insomnia: Wk 24 Missing | 0 | 0 | 4 | 0
  BL Clinical Insomnia, Moderate Severity: number analyzed (Participants) | 2 | 2 | 0 | 0
  BL Clinical Insomnia, Moderate Severity: Wk 24 No Clinically Significant Insomnia | 0 | 0 |  |
  BL Clinical Insomnia, Moderate Severity: Wk 24 Subthreshold Insomnia | 2 | 2 |  |
  BL Clinical Insomnia, Moderate Severity: Wk 24 Clinical Insomnia, Moderate Severity | 0 | 0 |  |
  BL Clinical Insomnia, Moderate Severity: Wk 24 Clinical Insomnia, Severe | 0 | 0 |  |
  BL Clinical Insomnia, Moderate Severity: Wk 24 Missing | 0 | 0 |  |
  BL Clinical Insomnia, Severe: number analyzed (Participants) | 0 | 0 | 0 | 0
  BL Clinical Insomnia, Severe: Wk 24 No Clinically Significant Insomnia |  | 0 |  |
  BL Missing: number analyzed (Participants) | 0 | 0 | 0 | 0

28. Secondary Outcome: Percentage of Participants Using Oral Rescue Therapy (ORT), Corticosteroid, or Bailout Rilonacept for Pericarditis Every 4 Weeks Cumulatively in the RW Period
Description: ORT included analgesics, NSAIDs, and/or colchicine. ORT use while waiting for at least 5 days since previous administration of study drug before receiving bailout, or within 5 days before the assessment of pericarditis recurrence, was excluded.
Time Frame: RW Period (mean 24.8 weeks)
Population: ITT Analysis Set: all participants who were randomized in the RW period.
Measure: Number; unit: percentage of participants
Arm/Group | Randomized Withdrawal Period: Rilonacept | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 30 | 31
percentage of participants
  ORT : First Use ≤ 4 Weeks | 0 | 3.2
  ORT : First Use ≤ 8 Weeks | 0 | 6.5
  ORT : First Use ≤ 12 Weeks | 0 | 6.5
  ORT : First Use ≤ 16 Weeks | 3.3 | 6.5
  ORT : First Use ≤ 20 Weeks | 3.3 | 6.5
  ORT : First Use ≤ 24 Weeks | 3.3 | 6.5
  ORT : All Weeks (Including > 24 Weeks in RW Period) | 3.3 | 6.5
  Corticosteroid : First Use ≤ 4 Weeks | 0 | 0
  Corticosteroid : First Use ≤ 8 Weeks | 0 | 0
  Corticosteroid : First Use ≤ 12 Weeks | 0 | 0
  Corticosteroid : First Use ≤ 16 Weeks | 0 | 0
  Corticosteroid : First Use ≤ 20 Weeks | 0 | 0
  Corticosteroid : First Use ≤ 24 Weeks | 0 | 0
  Corticosteroid : All Weeks (Including > 24 Weeks in RW Period) | 0 | 0
  Bailout : First Use ≤ 4 Weeks | 0 | 29.0
  Bailout : First Use ≤ 8 Weeks | 0 | 48.4
  Bailout : First Use ≤ 12 Weeks | 0 | 61.3
  Bailout : First Use ≤ 16 Weeks | 0 | 67.7
  Bailout : First Use ≤ 20 Weeks | 0 | 71.0
  Bailout : First Use ≤ 24 Weeks | 0 | 71.0
  Bailout : All Weeks (Including > 24 Weeks in RW Period) | 3.3 | 74.2
  Total (any of the above) : First Use ≤ 4 Weeks | 0 | 32.3
  Total (any of the above) : First Use ≤ 8 Weeks | 0 | 51.6
  Total (any of the above) : First Use ≤ 12 Weeks | 0 | 64.5
  Total (any of the above) : First Use ≤ 16 Weeks | 3.3 | 71.0
  Total (any of the above) : First Use ≤ 20 Weeks | 3.3 | 74.2
  Total (any of the above) : First Use ≤ 24 Weeks | 3.3 | 74.2
  Total (any of the above) : All Weeks (Including > 24 Weeks in RW Period) | 6.7 | 77.4
Statistical Analysis 1: Comparison: Randomized Withdrawal Period: Rilonacept vs Randomized Withdrawal Period: Placebo; Participants who used ORT, corticosteroids or bailout rilonacept during the RW Period; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Two-sided p value calculated using a Cochran-Mantel-Haenszel test adjudicated by randomization strata; Odds Ratio (OR) = 0.015, 95% CI 2-sided [0.002 to 0.108]

29. Secondary Outcome: Percentage of Participants Using ORT for Pericarditis in the First 24 Weeks of RW Period
Description: ORT included analgesics, NSAIDs, and/or colchicine.
Time Frame: RW Period (up to Week 24)
Population: ITT Analysis Set: all participants who were randomized in the RW period.
Measure: Number; unit: percentage of participants
Arm/Group | Randomized Withdrawal Period: Rilonacept | Randomized Withdrawal Period: Placebo
Number analyzed (Participants) | 30 | 31
percentage of participants | 3.3 | 6.5

30. Secondary Outcome: Percentage of Participants With Pericardial Delayed Hyperenhancement, Myocardial Delayed Hyperenhancement or Pericardial Effusion on Magnetic Resonance Imaging (MRI) at RW Week 24
Description: MRI assessments were performed in a subgroup of participants (MRI substudy) to assess the percentage of participants with:
  * Pericardial delayed hyperenhancement
  * Myocardial delayed hyperenhancement
  * Pericardial effusion
Time Frame: RW Period Week 24
Population: ITT Week 24 Analysis Set: All participants randomized at least 24 weeks before data cutoff. Participants in the MRI substudy with nonmissing data.
Measure: Number; unit: percentage of participants
Arm/Group | Randomized Withdrawal Period: Rilonacept, Before Bailout Rilonacept | Randomized Withdrawal Period: Rilonacept, Including Bailout Rilonacept | Randomized Withdrawal Period: Placebo | Randomized Withdrawal Period: Placebo, Including Bailout Rilonacept
Number analyzed (Participants) | 6 | 6 | 3 | 3
percentage of participants
  Pericardial Delayed Hyperenhancement | 66.7 | 66.7 | 28.6 | 57.1
  Myocardial Delayed Hyperenhancement | 0 | 0 | 0 | 0
  Pericardial Effusion | 0 | 0 | 0 | 0

31. Secondary Outcome: Time From First Dose to Pain Response in the RI Period
Description: Participants were asked to select the score that best described their average level of pericarditis pain over the previous 24 hours using an 11-point numerical rating scale (NRS), where zero (0) indicates 'no pain' and ten (10) indicates 'pain as bad as it could be'. Time to pain response was defined as number of days from first dose to the first day a participant's daily pain NRS was ≤ 2 of the 3 days over which the rolling average daily pain NRS was ≤ 2.
Time Frame: RI Period (up to 12 weeks)
Population: Run-in Analysis Set: All participants who received at least 1 dose of study drug in the RI period. Participants with a baseline NRS measurement >= 3.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Run-in Period: Single-blind rilonacept 320 mg (or 4.4 mg/kg in pediatric participants ≥ 12 and < 18 years old) subcutaneous (SC), followed by 160 mg (or 2.2 mg/kg in pediatric participants ≥12 and <18 years old) injections once weekly for 12 weeks.
Arm/Group | Run-in Period
Number analyzed (Participants) | 66
days | 5.0 [4.0 to 6.0]

32. Secondary Outcome: Time From First Dose to CRP Normalization in the RI Period
Description: Time to CRP normalization, defined as CRP ≤ 0.5 mg/dL, was censored at treatment discontinuation, taking prohibited medication, or Week 12, whichever occurred first.
Time Frame: RI Period (up to 12 weeks)
Population: Run-in Analysis Set: All participants who received at least 1 dose of study drug in the RI period. Participants with a baseline CRP measurement >= 0.5 mg/dL.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Run-in Period
Number analyzed (Participants) | 69
days | 7.0 [5.0 to 8.0]

33. Secondary Outcome: Time From First Dose to Rilonacept Monotherapy in RI Period
Description: Time to rilonacept monotherapy was defined as the number of weeks from first dose to the first day of achieving monotherapy.
Time Frame: RI Period (up to 12 weeks)
Population: Run-in Analysis Set: All participants who received at least 1 dose of study drug in the RI period. Participants with background therapies at RI Baseline.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Run-in Period
Number analyzed (Participants) | 79
weeks | 7.3 [7.0 to 8.1]

34. Secondary Outcome: Time From First Dose to Treatment Response in RI Period
Description: Time to treatment response is defined as time from first dose to the first day of pain response, and CRP ≤ 0.5 mg/dL within 7 days before or after pain response. Treatment response day will be the first day that the above criterion is met. If pain response occurs before CRP ≤ 0.5 mg/dL, each 3-day rolling average of NRS should be ≤ 2.0 from the day of pain response to the day of CRP ≤ 0.5 mg/dL. The response day will be the day of pain response. If CRP ≤0.5 mg/dL occurs before pain response, the response day will also be the day of pain response.
Time Frame: RI Period (up to 12 weeks)
Population: Run-in Analysis Set: All participants who received at least 1 dose of study drug in the RI period. Participants with baseline measurements of CRP >0.5 mg/dL and NRS > 2.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Run-in Period
Number analyzed (Participants) | 79
days | 5.0 [4.0 to 7.0]

35. Secondary Outcome: Percentage of Participants Achieving Clinical Response at RI Period Week 12
Description: Participants were asked to select the score that best described their average level of pericarditis pain over the previous 24 hours using an 11-point numerical rating scale (NRS), where zero (0) indicates 'no pain' and ten (10) indicates 'pain as bad as it could be'. Clinical Response was defined as a weekly average of daily pericarditis pain of ≤ 2.0 on the 11-point NRS and CRP level ≤ 0.5 mg/dL and participants must have been able to stop background SOC pericarditis therapy by Week 10.
Time Frame: RI Period Week 12
Population: Run-in Analysis Set: All participants who received at least 1 dose of study drug in the RI period. Participants achieving treatment response in the RI period.
Measure: Number; unit: percentage of participants
Arm/Group | Run-in Period
Number analyzed (Participants) | 86
percentage of participants
  Achieved Clinical Response | 84.9
  Did Not Achieve Clinical Response | 15.1

36. Secondary Outcome: Percentage of Participants With CRP Normalization at RI Period Week 12
Description: CRP normalization was defined as CRP ≤ 0.5 mg/dL.
Time Frame: RI Period Week 12
Population: Run-in Analysis Set: All participants who received at least 1 dose of study drug in the RI period. Participants with a baseline CRP measurement ≥ 0.5 mg/dL.
Measure: Number; unit: percentage of participants
Arm/Group | Run-in Period
Number analyzed (Participants) | 69
percentage of participants | 98.6

37. Secondary Outcome: Change From Baseline Over Time in Weekly Average of Pericarditis Pain NRS Score in RI Period
Description: as for outcome 12
Time Frame: RI Period Baseline, RI Period Weeks 1-12
Population: Run-in Analysis Set: All participants who received at least 1 dose of study drug in the RI period. Participants with an assessment at given time period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Run-in Period
Number analyzed (Participants) | 86
score on a scale
  RI Baseline: number analyzed (Participants) | 84
  RI Baseline | 4.48 (2.510)
  Change at RI Week 1: number analyzed (Participants) | 81
  Change at RI Week 1 | -2.31 (2.187)
  Change at RI Week 2: number analyzed (Participants) | 79
  Change at RI Week 2 | -3.18 (2.605)
  Change at RI Week 3: number analyzed (Participants) | 78
  Change at RI Week 3 | -3.28 (2.547)
  Change at RI Week 4: number analyzed (Participants) | 80
  Change at RI Week 4 | -3.51 (2.614)
  Change at RI Week 5: number analyzed (Participants) | 80
  Change at RI Week 5 | -3.55 (2.661)
  Change at RI Week 6: number analyzed (Participants) | 80
  Change at RI Week 6 | -3.70 (2.615)
  Change at RI Week 7: number analyzed (Participants) | 79
  Change at RI Week 7 | -3.81 (2.663)
  Change at RI Week 8: number analyzed (Participants) | 79
  Change at RI Week 8 | -3.92 (2.569)
  Change at RI Week 9: number analyzed (Participants) | 78
  Change at RI Week 9 | -3.81 (2.727)
  Change at RI Week 10: number analyzed (Participants) | 80
  Change at RI Week 10 | -3.83 (2.649)
  Change at RI Week 11: number analyzed (Participants) | 79
  Change at RI Week 11 | -4.05 (2.596)
  Change at RI Week 12: number analyzed (Participants) | 77
  Change at RI Week 12 | -4.00 (2.658)

38. Secondary Outcome: Change From Baseline Over Time in CRP Levels in RI Period
Time Frame: RI Period Baseline, RI Period Day 4, Weeks 1, 2, 4, 6, 12
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Run-in Period
Number analyzed (Participants) | 85
mg/dL
  RI Baseline | 3.72 (5.719)
  Change at RI Day 4: number analyzed (Participants) | 78
  Change at RI Day 4 | -2.80 (4.582)
  Change at RI Week 1: number analyzed (Participants) | 81
  Change at RI Week 1 | -3.48 (5.539)
  Change at RI Week 2: number analyzed (Participants) | 80
  Change at RI Week 2 | -3.55 (5.717)
  Change at RI Week 4: number analyzed (Participants) | 78
  Change at RI Week 4 | -3.46 (5.809)
  Change at RI Week 6: number analyzed (Participants) | 81
  Change at RI Week 6 | -3.55 (5.899)
  Change at RI Week 12: number analyzed (Participants) | 81
  Change at RI Week 12 | -3.60 (5.916)

39. Secondary Outcome: Percentage of Participants With Resolution of Pericarditis-Related ECHO and ECG Abnormalities at Week 12 of the RI Period
Time Frame: RI Period Baseline, RI Period Week 12
Population: Run-in Analysis Set: All participants who received at least 1 dose of study drug in the RI period. Participants with ECHO and ECG abnormalities at RI Baseline.
Measure: Number; unit: percentage of participants
Groups:
- Run-in Period: ECHO Abnormality at Baseline: Participants with an ECHO abnormality (ST-Elevation) at RI period baseline.
- Run-in Period: ECG Abnormality (ST-Elevation) at Baseline: Participants with an ECG abnormality (ST-elevation) at RI period baseline.
- Run-in Period: ECG Abnormality (PR Depression) at Baseline: Participants with an ECG abnormality (PR depression) at RI period baseline.
Arm/Group | Run-in Period: ECHO Abnormality at Baseline | Run-in Period: ECG Abnormality (ST-Elevation) at Baseline | Run-in Period: ECG Abnormality (PR Depression) at Baseline
Number analyzed (Participants) | 11 | 6 | 6
percentage of participants | 63.6 | 100 | 100

40. Secondary Outcome: Percentage of Days With No or Minimal Pain in the RI Period While on Treatment
Description: No or minimal pain is defined as non-missing daily NRS ≤ 2, where participants were asked to select the score that best describes their average level of pericarditis pain over the previous 24 hours using an 11-point NRS, where zero (0) indicates 'no pain' and ten (10) indicates 'pain as bad as it could be'.
Time Frame: RI Period (up to Week 12)
Population: Run-in Analysis Set: All participants who received at least 1 dose of study drug in the RI period.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Run-in Period
Number analyzed (Participants) | 86
percentage of days | 80.66 (21.388)

41. Secondary Outcome: Percentage of Participants With No or Minimal Pericarditis Symptoms Over Time in the RI Period, Based on the PGIPS
Description: as for outcome 20
Time Frame: RI Period Baseline, RI Period Weeks 6 and 12
Population: Run-in Analysis Set: All participants who received at least 1 dose of study drug in the RI period. Participants with an assessment at given time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Run-in Period
Number analyzed (Participants) | 83
percentage of participants
  Baseline | 18.1 [10.48 to 28.05]
  Week 6: number analyzed (Participants) | 76
  Week 6 | 89.5 [80.31 to 95.34]
  Week 12: number analyzed (Participants) | 81
  Week 12 | 92.6 [84.57 to 97.23]

42. Secondary Outcome: Percentage of Participants With No or Minimal Pericarditis Activity Over Time in the RI Period, Based on the PGA-PA
Description: The PGA-PA is a single-item, clinician-reported outcome measure that Investigators use to rate their impression of the patient's overall pericarditis disease activity at the time the assessment is completed, using a rating scale ranging from absent to very severe. The Investigator selected the box that best described a participant's pericarditis activity at the time of occurrence of the assessment: Absent, Minimal, Mild, Moderate, Moderately Severe, Severe, Very Severe.
  The exact 95% CI is calculated with randomization strata pooled. Participants who had received bailout rilonacept or rescue medication before the time point were considered nonresponders.
Time Frame: RI Period Baseline, RI Period Weeks 6 and 12
Population: as for outcome 41
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Run-in Period
Number analyzed (Participants) | 86
percentage of participants
  RI Baseline: number analyzed (Participants) | 85
  RI Baseline | 10.6 [4.96 to 19.15]
  RI Week 6: number analyzed (Participants) | 77
  RI Week 6 | 94.8 [87.23 to 98.57]
  RI Week 12: number analyzed (Participants) | 78
  RI Week 12 | 98.7 [93.06 to 99.97]

43. Secondary Outcome: Change From RI Period Baseline in the SF-36 Domain Scores and Physical and Mental Scores to RI Period Week 12
Description: as for outcome 23
Time Frame: RI Period Baseline, RI Period Week 12
Population: as for outcome 41
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Run-in Period
Number analyzed (Participants) | 71
score on a scale
  Physical Component Score | 13.8 (8.7)
  Mental Component Score | 9.2 (9.3)
  Physical Functioning | 10.1 (9.2)
  Role-Physical | 13.8 (9.4)
  Bodily Pain | 19.1 (10.3)
  General Health | 7.7 (8.2)
  Vitality | 13.4 (9.9)
  Social Functioning | 15.1 (10.6)
  Role-Emotional | 7.7 (10.0)
  Mental Health | 9.6 (9.0)

44. Secondary Outcome: Change From RI Period Baseline in SF-6D Scores at RI Period Week 12
Description: as for outcome 24
Time Frame: RI Period Baseline, RI Period Week 12
Population: Run-in Analysis Set: All participants who received at least 1 dose of study drug in the RI period. Participants with an assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Run-in Period
Number analyzed (Participants) | 71
score on a scale | 0.1828 (0.12658)

45. Secondary Outcome: Change From RI Period Baseline in 5-level EuroQoL-5 Dimensions (EQ-5D-5L) Individual Scores and Index Value at RI Period Week 12
Description: as for outcome 25
Time Frame: RI Period Baseline, RI Period Week 12
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Run-in Period
Number analyzed (Participants) | 74
score on a scale
  Mobility | -0.2 (0.84)
  Self-Care | -0.1 (0.57)
  Usual Activities | -1.1 (1.16)
  Pain/Discomfort | -1.5 (1.18)
  Anxiety/Depression | -0.5 (0.90)
  Index Score | 0.1626 (0.16814)
  VAS Score | 23.0 (23.41)

46. Secondary Outcome: Change From RI Period Baseline in ISI Total Score at RI Period Week 12
Description: as for outcome 26
Time Frame: RI Period Baseline, RI Period Week 12
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Run-in Period
Number analyzed (Participants) | 72
score on a scale | -4.9 (6.31)

47. Secondary Outcome: Change in ISI Categories From RI Period Baseline to RI Period Week 12
Description: as for outcome 26
Time Frame: RI Period Baseline (BL), RI Period Week (Wk) 12
Population: Run-in Analysis Set: All participants who received at least 1 dose of study drug in the RI period. Participants 18 years or older with an assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Period
Number analyzed (Participants) | 79
Participants
  BL No Clinically Significant Insomnia: number analyzed (Participants) | 26
  BL No Clinically Significant Insomnia: Wk 12 No Clinically Significant Insomnia | 23
  BL No Clinically Significant Insomnia: Wk 12 Subthreshold Insomnia | 1
  BL No Clinically Significant Insomnia: Wk 12 Clinical Insomnia, Moderate Severity | 1
  BL No Clinically Significant Insomnia: Wk 12 Clinical Insomnia, Severe | 0
  BL No Clinically Significant Insomnia: Wk 12 Missing | 1
  BL Subthreshold Insomnia: number analyzed (Participants) | 27
  BL Subthreshold Insomnia: Wk 12 No Clinically Significant Insomnia | 18
  BL Subthreshold Insomnia: Wk 12 Subthreshold Insomnia | 7
  BL Subthreshold Insomnia: Wk 12 Clinical Insomnia, Moderate Severity | 0
  BL Subthreshold Insomnia: Wk 12 Clinical Insomnia, Severe | 0
  BL Subthreshold Insomnia: Wk 12 Missing | 2
  BL Clinical Insomnia, Moderate Severity: number analyzed (Participants) | 19
  BL Clinical Insomnia, Moderate Severity: Wk 12 No Clinically Significant Insomnia | 7
  BL Clinical Insomnia, Moderate Severity: Wk 12 Subthreshold Insomnia | 10
  BL Clinical Insomnia, Moderate Severity: Wk 12 Clinical Insomnia, Moderate Severity | 2
  BL Clinical Insomnia, Moderate Severity: Wk 12 Clinical Insomnia, Severe | 0
  BL Clinical Insomnia, Moderate Severity: Wk 12 Missing | 0
  BL Clinical Insomnia, Severe: number analyzed (Participants) | 4
  BL Clinical Insomnia, Severe: Wk 12 No Clinically Significant Insomnia | 2
  BL Clinical Insomnia, Severe: Wk 12 Subthreshold Insomnia | 0
  BL Clinical Insomnia, Severe: Wk 12 Clinical Insomnia, Moderate Severity | 1
  BL Clinical Insomnia, Severe: Wk 12 Clinical Insomnia, Severe | 0
  BL Clinical Insomnia, Severe: Wk 12 Missing | 1
  BL Missing: number analyzed (Participants) | 3
  BL Missing: Wk 12 No Clinically Significant Insomnia | 3
  BL Missing: Wk 12 Subthreshold Insomnia | 0
  BL Missing: Wk 12 Clinical Insomnia, Moderate Severity | 0
  BL Missing: Wk 12 Clinical Insomnia, Severe | 0
  BL Missing: Wk 12 Missing | 0

48. Secondary Outcome: Number of Participants Who Were Off Background Pericarditis Medication on or Before RI Period Weeks 4, 8, 10, and 12
Time Frame: RI Period Baseline, RI Period Weeks 4, 8, 10, 12
Population: Run-in Analysis Set: All participants who received at least 1 dose of study drug in the RI period. Participants 18 years or older with an assessment at given time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Period
Number analyzed (Participants) | 86
Participants
  RI Baseline: Not Receiving Background Pericarditis Medication | 7
  RI Baseline: Receiving Background Pericarditis Medication | 79
  RI Week 4: number analyzed (Participants) | 84
  RI Week 4: Not Receiving Background Pericarditis Medication | 15
  RI Week 4: Receiving Background Pericarditis Medication | 69
  RI Week 8: number analyzed (Participants) | 81
  RI Week 8: Not Receiving Background Pericarditis Medication | 49
  RI Week 8: Receiving Background Pericarditis Medication | 32
  RI Week 10: number analyzed (Participants) | 80
  RI Week 10: Not Receiving Background Pericarditis Medication | 71
  RI Week 10: Receiving Background Pericarditis Medication | 9
  RI Week 12: number analyzed (Participants) | 79
  RI Week 12: Not Receiving Background Pericarditis Medication | 76
  RI Week 12: Receiving Background Pericarditis Medication | 3

49. Secondary Outcome: Annualized Rate of Pericarditis Recurrence in the Long-Term Extension (LTE) Period Based on Investigator's Assessment (Based on Investigators' Judgement)
Description: Annualized Recurrence Rate is defined as the number of recurrences in LTE periods for all participants/Sum of participant years in LTE periods for all participants. Participant years in LTE period is defined as the time from 1st dose date of LTE period to the date of End of Study, or data cutoff date, whichever is earlier. The 95% CI was calculated using an exact method with Poisson distribution. Pericarditis recurrence is defined as the recurrence of typical pericarditis pain associated with supportive objective evidence of pericarditis.
Time Frame: LTE Period, through LTE Follow up (up to Week 48)
Population: LTE Analysis Set: participants who consented to LTE period and took at least 1 dose of study drug in the LTE period.
Measure: Number (95% Confidence Interval); unit: recurrences per participant per year
Groups:
- Long Term Extension: Overall: All participants who entered the LTE and received up to 24 months of open-label rilonacept 160 mg (or 2.2 mg/kg for pediatric participants) SC injections once weekly based on their clinical status and at the discretion of the Investigator.
Arm/Group | Long Term Extension: Non-Randomized | Long Term Extension: Randomized, Recurrence (RW) | Long Term Extension: Randomized, No Recurrence (RW) | Long Term Extension: Overall
Number analyzed (Participants) | 15 | 25 | 34 | 74
recurrences per participant per year | 0.088 [0.011 to 0.319] | 0.168 [0.062 to 0.367] | 0.125 [0.046 to 0.273] | 0.132 [0.072 to 0.221]

50. Secondary Outcome: Change From LTE Baseline Over Time in CRP Levels
Time Frame: LTE Baseline, LTE Week 12, LTE Week 24
Population: Long term extension (LTE) Analysis Set: participants who consented to LTE period and took at least 1 dose of study drug in the LTE period. Participants with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Long Term Extension: Non-Randomized: Participants who entered the LTE directly from RI after protocol-specified 22 adjudicated pericarditis recurrence events had accrued.
- Long Term Extension: Randomized, Recurrence (RW): Participants who consented to LTE period and took at least 1 dose of study drug in the LTE period.
  Participants with recurrence as evaluated based on CEC adjudication in Randomization Withdrawal period.
- Long Term Extension: Randomized, No Recurrence (RW): Participants who consented to LTE period and took at least 1 dose of study drug in the LTE period.
  Participants with no recurrence as evaluated based on CEC adjudication in Randomization Withdrawal period.
Arm/Group | Long Term Extension: Non-Randomized | Long Term Extension: Randomized, Recurrence (RW) | Long Term Extension: Randomized, No Recurrence (RW) | Long Term Extension: Overall
Number analyzed (Participants) | 15 | 25 | 34 | 74
mg/dL
  LTE Baseline | 0.18 (0.294) | 0.21 (0.249) | 0.16 (0.251) | 0.18 (0.257)
  Change at Week 12: number analyzed (Participants) | 15 | 24 | 33 | 72
  Change at Week 12 | 0.01 (0.249) | 0.00 (0.127) | -0.06 (0.255) | -0.03 (0.219)
  Change at Week 24: number analyzed (Participants) | 14 | 25 | 31 | 70
  Change at Week 24 | 0.03 (0.182) | 0.17 (0.909) | -0.06 (0.269) | 0.04 (0.579)

51. Secondary Outcome: Percentage of Participants With Absent or Minimal Pericarditis Activity In the LTE Period Based on the PGIPS
Description: Percentage of participants with no or minimal pericarditis symptoms in the LTE Period, based on the PGIPS, a single-item measure of the participant's impression of the overall severity of pericarditis symptoms at the time the questionnaire is administered using a 7-point rating scale ranging from absent (0=no recurrent pericarditis symptoms) to very severe (6=recurrent pericarditis symptoms that cannot be ignored and markedly limits daily activities).
Time Frame: LTE Baseline, LTE Month 12, LTE Month 24
Population: as for outcome 50
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Long Term Extension: Non-Randomized | Long Term Extension: Randomized, Recurrence (RW) | Long Term Extension: Randomized, No Recurrence (RW) | Long Term Extension: Overall
Number analyzed (Participants) | 15 | 25 | 34 | 74
percentage of participants
  LTE Baseline | 100.0 [78.20 to 100.0] | 88.0 [68.78 to 97.45] | 91.2 [76.32 to 98.14] | 91.9 [83.18 to 96.97]
  LTE Week 12: number analyzed (Participants) | 15 | 24 | 32 | 71
  LTE Week 12 | 93.3 [68.05 to 99.83] | 95.8 [78.88 to 99.89] | 100.0 [89.11 to 100.00] | 97.2 [90.19 to 99.66]
  LTE Week 24: number analyzed (Participants) | 15 | 23 | 30 | 68
  LTE Week 24 | 86.7 [59.54 to 98.34] | 78.3 [56.30 to 92.54] | 93.3 [77.93 to 99.18] | 86.8 [76.36 to 93.77]

52. Secondary Outcome: Percentage of Participants With Absent or Minimal Pericarditis Activity Over Time in the LTE Period Based on the PGA-PA
Description: as for outcome 21
Time Frame: LTE Baseline, LTE Week 12, LTE Week 24
Population: as for outcome 50
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Long-Term Extension: Overall: All participants who entered the LTE and received up to 24 months of open-label rilonacept 160 mg (or 2.2 mg/kg for pediatric participants) SC injections once weekly based on their clinical status and at the discretion of the Investigator.
Arm/Group | Long Term Extension: Non-Randomized | Long Term Extension: Randomized, Recurrence (RW) | Long Term Extension: Randomized, No Recurrence (RW) | Long-Term Extension: Overall
Number analyzed (Participants) | 15 | 25 | 34 | 74
percentage of participants
  LTE Baseline | 100.0 [78.20 to 100.0] | 92.0 [73.97 to 99.02] | 94.1 [80.32 to 99.28] | 94.6 [86.73 to 98.51]
  LTE Week 12: number analyzed (Participants) | 15 | 24 | 33 | 72
  LTE Week 12 | 100.0 [78.20 to 100.00] | 91.7 [73.00 to 98.97] | 97.0 [84.24 to 99.92] | 95.8 [88.30 to 99.13]
  LTE Week 24: number analyzed (Participants) | 15 | 25 | 31 | 71
  LTE Week 24 | 93.3 [68.05 to 99.83] | 88.0 [68.78 to 97.45] | 96.8 [83.30 to 99.92] | 93.0 [84.33 to 97.67]

53. Secondary Outcome: Change From LTE Baseline in the SF-36 Domain Scores and Physical and Mental Scores
Description: as for outcome 23
Time Frame: LTE Baseline, LTE Week 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Long Term Extension: Non-Randomized | Long Term Extension: Randomized, Recurrence (RW) | Long Term Extension: Randomized, No Recurrence (RW) | Long-Term Extension: Overall
Number analyzed (Participants) | 14 | 23 | 29 | 66
score on a scale
  Physical Functioning: Change at LTE Week 24 | 2.596 (8.4132) | 0.125 (6.4017) | -0.463 (5.7067) | 0.391 (6.5919)
  Role-Physical: Change at LTE Week 24 | -1.443 (6.0141) | 2.052 (9.8327) | -1.627 (6.6000) | -0.306 (7.8579)
  Bodily Pain: Change at LTE Week 24 | 3.082 (10.2083) | 1.140 (9.6306) | -0.820 (8.0536) | 0.690 (9.0827)
  General Health: Change at LTE Week 24 | 1.324 (10.1092) | 0.932 (7.0108) | 0.762 (6.1724) | 0.940 (7.3166)
  Vitality: Change at LTE Week 24 | 1.910 (8.2069) | 1.679 (9.3889) | -0.307 (6.6591) | 0.855 (7.9681)
  Social Functioning: Change at LTE Week 24 | -0.716 (7.8320) | 0.219 (10.0797) | 0.172 (6.4927) | 0.000 (8.0595)
  Role-Emotional: Change at LTE Week 24 | 0.496 (6.3849) | 0.758 (5.6497) | -0.360 (8.0771) | 0.211 (6.8796)
  Mental Health: Change at LTE Week 24 | 2.988 (9.8321) | 0.455 (8.2976) | 1.353 (8.2616) | 1.387 (8.5381)
  Physical Score: Change at LTE Week 24 | 1.210 (6.5951) | 1.168 (8.0082) | -1.079 (6.3170) | 0.190 (6.9912)
  Mental Score: Change at LTE Week 24 | 1.186 (7.5539) | 0.596 (6.6219) | 0.850 (8.8099) | 0.833 (7.7298)

54. Secondary Outcome: Change From LTE Baseline in SF-6D Health Utility Index Score
Description: The SF-6D is calculated based on responses to 11 items on the SF-36, that correspond to 6 domains: physical functioning, role participation (combined role-physical and role-emotional), social functioning, bodily pain, mental health, and vitality. Individual respondents can be classified on any of 4 to 6 levels of functioning or limitations for each of six domains, thus allowing a respondent to be classified into any of 18,000 possible unique health states. Using a standard gamble technique, each of these health states were mapped onto the SF-6D index score, which ranges from 0.00 (worst possible health state/death) to 1.00 (best possible health state/perfect health).
Time Frame: LTE Baseline, LTE Week 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Long Term Extension: Non-Randomized | Long Term Extension: Randomized, Recurrence (RW) | Long Term Extension: Randomized, No Recurrence (RW) | Long Term Extension: Overall
Number analyzed (Participants) | 14 | 23 | 29 | 66
score on a scale | -0.106 (0.4449) | 0.163 (0.4368) | 0.003 (0.0781) | 0.035 (0.3425)

55. Secondary Outcome: Change From LTE Baseline in EQ-5D-5L Individual Scores and Index Value
Description: as for outcome 25
Time Frame: LTE Baseline, LTE Week 24
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Long Term Extension: Non-Randomized | Long Term Extension: Randomized, Recurrence (RW) | Long Term Extension: Randomized, No Recurrence (RW) | Long-Term Extension: Overall
Number analyzed (Participants) | 14 | 23 | 30 | 67
score on a scale
  Mobility: Change at LTE Week 24 | -0.2 (0.70) | 0.0 (0.77) | 0.1 (0.48) | 0.0 (0.64)
  Self-Care: Change at LTE Week 24 | 0.1 (1.00) | -0.1 (0.29) | 0.0 (0.18) | 0.0 (0.49)
  Usual Activities: Change at LTE Week 24 | -0.1 (1.35) | 0.0 (0.80) | -0.1 (0.45) | -0.1 (0.81)
  Pain/Discomfort: Change at Week 24 | -0.3 (1.20) | -0.2 (0.85) | 0.0 (0.67) | -0.1 (0.86)
  Anxiety/Depression: Change at Week 24 | -0.1 (0.73) | 0.1 (0.67) | 0.0 (0.72) | 0.0 (0.70)
  Index Score: Change at Week 24 | 0.0546 (0.19544) | 0.0290 (0.10339) | -0.0004 (0.10212) | 0.0212 (0.12704)
  VAS Score: Change at Week 24 | 6.2 (25.95) | 12.6 (27.07) | -0.2 (9.48) | 5.5 (21.19)

56. Secondary Outcome: Change From LTE Baseline in ISI Total Score
Description: as for outcome 26
Time Frame: LTE Baseline, LTE Week 24
Population: Long term extension (LTE) Analysis Set: participants who consented to LTE period and took at least 1 dose of study drug in the LTE period. Participants 18 years or older with an assessment at given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Long Term Extension: Non-Randomized | Long Term Extension: Randomized, Recurrence (RW) | Long Term Extension: Randomized, No Recurrence (RW) | Long-Term Extension: Overall
Number analyzed (Participants) | 12 | 22 | 29 | 63
score on a scale | -0.3 (1.87) | -0.2 (6.87) | -1.1 (3.58) | -0.1 (0.89)

57. Secondary Outcome: Change From LTE Baseline in ISI Categories
Description: as for outcome 26
Time Frame: LTE Baseline (BL), LTE Week 24
Population: as for outcome 56
Measure: Count of Participants; unit: Participants
Arm/Group | Long Term Extension: Non-Randomized | Long Term Extension: Randomized, Recurrence (RW) | Long Term Extension: Randomized, No Recurrence (RW) | Long-Term Extension: Overall
Number analyzed (Participants) | 12 | 24 | 32 | 68
Participants
  LTE BL No Clinically Significant Insomnia: number analyzed (Participants) | 10 | 14 | 23 | 47
  LTE BL No Clinically Significant Insomnia: LTE Week 24 No Clinically Significant Insomnia | 9 | 11 | 18 | 38
  LTE BL No Clinically Significant Insomnia: LTE Week 24 Subthreshold Insomnia | 1 | 2 | 4 | 7
  LTE BL No Clinically Significant Insomnia: LTE Week 24 Clinical Insomnia (Moderate Severity) | 0 | 0 | 0 | 0
  LTE BL No Clinically Significant Insomnia: LTE Week 24 Clinical Insomnia (Severe) | 0 | 1 | 0 | 1
  LTE BL No Clinically Significant Insomnia: LTE Week 24 Missing | 0 | 0 | 1 | 1
  LTE BL Subthreshold Insomnia: number analyzed (Participants) | 2 | 6 | 6 | 14
  LTE BL Subthreshold Insomnia: LTE Week 24 No Clinically Significant Insomnia | 0 | 2 | 3 | 5
  LTE BL Subthreshold Insomnia: LTE Week 24 Subthreshold Insomnia | 2 | 2 | 2 | 6
  LTE BL Subthreshold Insomnia: LTE Week 24 Clinical Insomnia (Moderate Severity) | 0 | 1 | 0 | 1
  LTE BL Subthreshold Insomnia: LTE Week 24 Clinical Insomnia (Severe) | 0 | 0 | 0 | 0
  LTE BL Subthreshold Insomnia: LTE Week 24 Missing | 0 | 1 | 1 | 2
  LTE BL Clinical Insomnia (Moderate Severity): number analyzed (Participants) | 0 | 3 | 3 | 6
  LTE BL Clinical Insomnia (Moderate Severity): LTE Week 24 No Clinically Significant Insomnia | 0 | 1 | 1 | 2
  LTE BL Clinical Insomnia (Moderate Severity): LTE Week 24 Subthreshold Insomnia | 0 | 2 | 0 | 2
  LTE BL Clinical Insomnia (Moderate Severity): LTE Week 24 Clinical Insomnia (Moderate Severity) | 0 | 0 | 1 | 1
  LTE BL Clinical Insomnia (Moderate Severity): LTE Week 24 Clinical Insomnia (Severe) | 0 | 0 | 0 | 0
  LTE BL Clinical Insomnia (Moderate Severity): LTE Week 24 Missing | 0 | 0 | 1 | 1
  LTE BL Clinical Insomnia (Severe): number analyzed (Participants) | 0 | 1 | 0 | 1
  LTE BL Clinical Insomnia (Severe): LTE Week 24 No Clinically Significant Insomnia | 0 | 0 | 0 | 0
  LTE BL Clinical Insomnia (Severe): LTE Week 24 Subthreshold Insomnia | 0 | 0 | 0 | 0
  LTE BL Clinical Insomnia (Severe): LTE Week 24 Clinical Insomnia (Moderate Severity) | 0 | 0 | 0 | 0
  LTE BL Clinical Insomnia (Severe): LTE Week 24 Clinical Insomnia (Severe) | 0 | 0 | 0 | 0
  LTE BL Clinical Insomnia (Severe): LTE Week 24 Missing | 0 | 1 | 0 | 1
  LTE BL Missing: number analyzed (Participants) | 0 | 0 | 0 | 0
  LTE BL Missing: LTE Week 24 No Clinically Significant Insomnia | 0 | 0 | 0 | 0
  LTE BL Missing: LTE Week 24 Subthreshold Insomnia | 0 | 0 | 0 | 0
  LTE BL Missing: LTE Week 24 Clinical Insomnia (Moderate Severity) | 0 | 0 | 0 | 0
  LTE BL Missing: LTE Week 24 Clinical Insomnia (Severe) | 0 | 0 | 0 | 0
  LTE BL Missing: LTE Week 24 Missing | 0 | 0 | 0 | 0

58. Secondary Outcome: Percentage of Participants Requiring Addition of Standard of Care (SOC) Pericarditis Therapy Every 4 Weeks Cumulatively in the LTE Period
Time Frame: LTE Period, through LTE Follow up (up to Week 24)
Population: This analysis was not done because Standard of Care treatment was not initiated in the LTE period.
Arm/Group | Long Term Extension: Non-Randomized | Long Term Extension: Randomized, Recurrence (RW) | Long Term Extension: Randomized, No Recurrence (RW)
Number analyzed (Participants) | 0 | 0 | 0

59. Secondary Outcome: Change From LTE Baseline in Pericardial Signs in ECHO
Time Frame: LTE Baseline, LTE Week 24
Population: as for outcome 56
Measure: Count of Participants; unit: Participants
Arm/Group | Long Term Extension: Non-Randomized | Long Term Extension: Randomized, Recurrence (RW) | Long Term Extension: Randomized, No Recurrence (RW) | Long-Term Extension: Overall
Number analyzed (Participants) | 15 | 24 | 24 | 63
Participants
  No Change | 3 | 4 | 7 | 14
  New | 0 | 0 | 1 | 1
  Improving | 1 | 0 | 1 | 2
  Resolved | 0 | 1 | 1 | 2
  Missing | 3 | 2 | 0 | 5
  Not Applicable | 8 | 17 | 14 | 39

60. Secondary Outcome: Change From LTE Baseline in Pericardial Signs in ECG
Time Frame: LTE Baseline, LTE Week 24
Population: as for outcome 50
Measure: Count of Participants; unit: Participants
Arm/Group | Long Term Extension: Non-Randomized | Long Term Extension: Randomized, Recurrence (RW) | Long Term Extension: Randomized, No Recurrence (RW) | Long-Term Extension: Overall
Number analyzed (Participants) | 15 | 25 | 34 | 74
Participants
  LTE Baseline: Normal | 7 | 16 | 21 | 44
  LTE Baseline: Abnormal-Consistent With Pericarditis | 0 | 1 | 1 | 2
  LTE Baseline: Abnormal-Not Consistent With Pericarditis But Clinically Significant | 0 | 0 | 1 | 1
  LTE Baseline: Abnormal-Not Consistent With Pericarditis But Not Clinically Significant | 8 | 8 | 11 | 27
  LTE Week 24: number analyzed (Participants) | 15 | 25 | 31 | 71
  LTE Week 24: Normal | 8 | 15 | 19 | 42
  LTE Week 24: Abnormal-Consistent With Pericarditis | 0 | 1 | 1 | 2
  LTE Week 24: Abnormal-Not Consistent With Pericarditis But Clinically Significant | 1 | 0 | 2 | 3
  LTE Week 24: Abnormal-Not Consistent With Pericarditis But Not Clinically Significant | 6 | 9 | 9 | 24

61. Secondary Outcome: Change From LTE Baseline in Pericardial Signs in MRI
Time Frame: LTE Baseline, LTE Week 24
Population: LTE Analysis Set - Participants in MRI Substudy. The number analyzed on each row pertains to the number of participants with a given baseline status.
Measure: Number; unit: participants
Arm/Group | Long Term Extension: Non-Randomized | Long Term Extension: Randomized, Recurrence (RW) | Long Term Extension: Randomized, No Recurrence (RW) | Long Term Extension: Overall
Number analyzed (Participants) | 8 | 13 | 16 | 37
participants
  Pericardial Delayed Hyperenhancement Baseline Yes -> Week 24 Yes: number analyzed (Participants) | 4 | 9 | 10 | 23
  Pericardial Delayed Hyperenhancement Baseline Yes -> Week 24 Yes | 2 | 5 | 2 | 9
  Pericardial Delayed Hyperenhancement Baseline Yes -> Week 24 No: number analyzed (Participants) | 4 | 9 | 10 | 23
  Pericardial Delayed Hyperenhancement Baseline Yes -> Week 24 No | 1 | 1 | 0 | 2
  Pericardial Delayed Hyperenhancement Baseline Yes -> Week 24 Not Done: number analyzed (Participants) | 4 | 9 | 10 | 23
  Pericardial Delayed Hyperenhancement Baseline Yes -> Week 24 Not Done | 1 | 3 | 8 | 12
  Pericardial Delayed Hyperenhancement Baseline No -> Week 24 Yes: number analyzed (Participants) | 0 | 2 | 4 | 6
  Pericardial Delayed Hyperenhancement Baseline No -> Week 24 Yes |  | 0 | 0 | 0
  Pericardial Delayed Hyperenhancement Baseline No -> Week 24 No: number analyzed (Participants) | 0 | 2 | 4 | 6
  Pericardial Delayed Hyperenhancement Baseline No -> Week 24 No |  | 1 | 2 | 3
  Pericardial Delayed Hyperenhancement Baseline No -> Week 24 Not Done: number analyzed (Participants) | 0 | 2 | 4 | 6
  Pericardial Delayed Hyperenhancement Baseline No -> Week 24 Not Done |  | 1 | 2 | 3
  Pericardial Delayed Hyperenhancement Baseline Missing -> Week 24 Yes: number analyzed (Participants) | 4 | 2 | 2 | 8
  Pericardial Delayed Hyperenhancement Baseline Missing -> Week 24 Yes | 0 | 0 | 0 | 0
  Pericardial Delayed Hyperenhancement Baseline Missing -> Week 24 No: number analyzed (Participants) | 4 | 2 | 2 | 8
  Pericardial Delayed Hyperenhancement Baseline Missing -> Week 24 No | 0 | 1 | 0 | 1
  Pericardial Delayed Hyperenhancement Baseline Missing -> Week 24 Not Done: number analyzed (Participants) | 4 | 2 | 2 | 8
  Pericardial Delayed Hyperenhancement Baseline Missing -> Week 24 Not Done | 4 | 1 | 2 | 7
  Myocardial Delayed Hyperenhancement Baseline Yes -> Week 24 Yes: number analyzed (Participants) | 2 | 2 | 3 | 7
  Myocardial Delayed Hyperenhancement Baseline Yes -> Week 24 Yes | 0 | 0 | 0 | 0
  Myocardial Delayed Hyperenhancement Baseline Yes -> Week 24 No: number analyzed (Participants) | 2 | 2 | 3 | 7
  Myocardial Delayed Hyperenhancement Baseline Yes -> Week 24 No | 1 | 0 | 2 | 3
  Myocardial Delayed Hyperenhancement Baseline Yes -> Week 24 Not Done: number analyzed (Participants) | 2 | 2 | 3 | 7
  Myocardial Delayed Hyperenhancement Baseline Yes -> Week 24 Not Done | 1 | 2 | 1 | 4
  Myocardial Delayed Hyperenhancement Baseline No -> Week 24 Yes: number analyzed (Participants) | 2 | 9 | 11 | 22
  Myocardial Delayed Hyperenhancement Baseline No -> Week 24 Yes | 0 | 0 | 1 | 1
  Myocardial Delayed Hyperenhancement Baseline No -> Week 24 No: number analyzed (Participants) | 2 | 9 | 11 | 22
  Myocardial Delayed Hyperenhancement Baseline No -> Week 24 No | 2 | 6 | 1 | 9
  Myocardial Delayed Hyperenhancement Baseline No -> Week 24 Not Done: number analyzed (Participants) | 2 | 9 | 11 | 22
  Myocardial Delayed Hyperenhancement Baseline No -> Week 24 Not Done | 0 | 3 | 9 | 12
  Myocardial Delayed Hyperenhancement Baseline Missing -> Week 24 Yes: number analyzed (Participants) | 4 | 2 | 2 | 8
  Myocardial Delayed Hyperenhancement Baseline Missing -> Week 24 Yes | 0 | 0 | 0 | 0
  Myocardial Delayed Hyperenhancement Baseline Missing -> Week 24 No: number analyzed (Participants) | 4 | 2 | 2 | 8
  Myocardial Delayed Hyperenhancement Baseline Missing -> Week 24 No | 0 | 1 | 0 | 1
  Myocardial Delayed Hyperenhancement Baseline Missing -> Week 24 Not Done: number analyzed (Participants) | 4 | 2 | 2 | 8
  Myocardial Delayed Hyperenhancement Baseline Missing -> Week 24 Not Done | 4 | 1 | 2 | 7
  Pericardial Effusion Baseline Yes -> Week 24 Yes: number analyzed (Participants) | 1 | 1 | 0 | 2
  Pericardial Effusion Baseline Yes -> Week 24 Yes | 0 | 0 |  | 0
  Pericardial Effusion Baseline Yes -> Week 24 No: number analyzed (Participants) | 1 | 1 | 0 | 2
  Pericardial Effusion Baseline Yes -> Week 24 No | 1 | 1 |  | 2
  Pericardial Effusion Baseline Yes -> Week 24 Not Done: number analyzed (Participants) | 1 | 1 | 0 | 2
  Pericardial Effusion Baseline Yes -> Week 24 Not Done | 0 | 0 |  | 0
  Pericardial Effusion Baseline No -> Week 24 Yes: number analyzed (Participants) | 3 | 10 | 14 | 27
  Pericardial Effusion Baseline No -> Week 24 Yes | 0 | 0 | 0 | 0
  Pericardial Effusion Baseline No -> Week 24 No: number analyzed (Participants) | 3 | 10 | 14 | 27
  Pericardial Effusion Baseline No -> Week 24 No | 3 | 6 | 4 | 13
  Pericardial Effusion Baseline No -> Week 24 Not Done: number analyzed (Participants) | 3 | 10 | 14 | 27
  Pericardial Effusion Baseline No -> Week 24 Not Done | 0 | 4 | 10 | 14
  Pericardial Effusion Baseline Missing -> Week 24 Yes: number analyzed (Participants) | 4 | 2 | 2 | 8
  Pericardial Effusion Baseline Missing -> Week 24 Yes | 0 | 0 | 0 | 0
  Pericardial Effusion Baseline Missing -> Week 24 No: number analyzed (Participants) | 4 | 2 | 2 | 8
  Pericardial Effusion Baseline Missing -> Week 24 No | 0 | 1 | 0 | 1
  Pericardial Effusion Baseline Missing -> Week 24 Not Done: number analyzed (Participants) | 4 | 2 | 2 | 8
  Pericardial Effusion Baseline Missing -> Week 24 Not Done | 4 | 1 | 2 | 7

62. Secondary Outcome: Number of Participants With Pericardial Delayed Hyperenhancement, Myocardial Delayed Hyperenhancement or Pericardial Effusion at LTE Period Week 24
Time Frame: LTE Week 24
Population: Long term extension (LTE) Analysis Set - MRI Substudy: participants in MRI Substudy who consented to LTE period and took at least 1 dose of study drug in the LTE period. Participants 18 years or older with an assessment at given time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Long Term Extension: Non-Randomized | Long Term Extension: Randomized, Recurrence (RW) | Long Term Extension: Randomized, No Recurrence (RW) | Long Term Extension: Overall
Number analyzed (Participants) | 8 | 13 | 16 | 37
Participants
  LTE BL: Pericardial Delayed Hyperenhancement=Yes: number analyzed (Participants) | 4 | 9 | 10 | 23
  LTE BL: Pericardial Delayed Hyperenhancement=Yes: LTE Week 24=Yes | 2 | 5 | 2 | 9
  LTE BL: Pericardial Delayed Hyperenhancement=Yes: LTE Week 24=No | 1 | 1 | 0 | 2
  LTE BL: Pericardial Delayed Hyperenhancement=Yes: LTE Week 24=Missing | 1 | 3 | 8 | 12
  LTE BL: Pericardial Delayed Hyperenhancement=No: number analyzed (Participants) | 0 | 2 | 4 | 6
  LTE BL: Pericardial Delayed Hyperenhancement=No: LTE Week 24=Yes |  | 0 | 0 | 0
  LTE BL: Pericardial Delayed Hyperenhancement=No: LTE Week 24=No |  | 1 | 2 | 3
  LTE BL: Pericardial Delayed Hyperenhancement=No: LTE Week 24=Missing |  | 1 | 2 | 3
  LTE BL: Pericardial Delayed Hyperenhancement=Missing: number analyzed (Participants) | 4 | 2 | 2 | 8
  LTE BL: Pericardial Delayed Hyperenhancement=Missing: LTE Week 24=Yes | 0 | 0 | 0 | 0
  LTE BL: Pericardial Delayed Hyperenhancement=Missing: LTE Week 24=No | 0 | 1 | 0 | 1
  LTE BL: Pericardial Delayed Hyperenhancement=Missing: LTE Week 24=Missing | 4 | 1 | 2 | 7
  LTE BL: Myocardial Delayed Hyperenhancement=Yes: number analyzed (Participants) | 2 | 2 | 3 | 7
  LTE BL: Myocardial Delayed Hyperenhancement=Yes: LTE Week 24=Yes | 0 | 0 | 0 | 0
  LTE BL: Myocardial Delayed Hyperenhancement=Yes: LTE Week 24=No | 1 | 0 | 2 | 3
  LTE BL: Myocardial Delayed Hyperenhancement=Yes: LTE Week 24=Missing | 1 | 2 | 1 | 4
  LTE BL: Myocardial Delayed Hyperenhancement=No: number analyzed (Participants) | 2 | 9 | 11 | 22
  LTE BL: Myocardial Delayed Hyperenhancement=No: LTE Week 24=Yes | 0 | 0 | 1 | 1
  LTE BL: Myocardial Delayed Hyperenhancement=No: LTE Week 24=No | 2 | 6 | 1 | 9
  LTE BL: Myocardial Delayed Hyperenhancement=No: LTE Week 24=Missing | 0 | 3 | 9 | 12
  LTE BL: Myocardial Delayed Hyperenhancement=Missing: number analyzed (Participants) | 4 | 2 | 2 | 8
  LTE BL: Myocardial Delayed Hyperenhancement=Missing: LTE Week 24=Yes | 0 | 0 | 0 | 0
  LTE BL: Myocardial Delayed Hyperenhancement=Missing: LTE Week 24=No | 0 | 1 | 0 | 1
  LTE BL: Myocardial Delayed Hyperenhancement=Missing: LTE Week 24=Missing | 4 | 1 | 2 | 7
  LTE BL: Pericardial Effusion=Yes: number analyzed (Participants) | 1 | 1 | 0 | 2
  LTE BL: Pericardial Effusion=Yes: LTE Week 24=Yes | 0 | 0 |  | 0
  LTE BL: Pericardial Effusion=Yes: LTE Week 24=No | 1 | 1 |  | 2
  LTE BL: Pericardial Effusion=Yes: LTE Week 24=Missing | 0 | 0 |  | 0
  LTE BL: Pericardial Effusion=No: number analyzed (Participants) | 3 | 10 | 14 | 27
  LTE BL: Pericardial Effusion=No: LTE Week 24=Yes | 0 | 0 | 0 | 0
  LTE BL: Pericardial Effusion=No: LTE Week 24=No | 3 | 6 | 4 | 13
  LTE BL: Pericardial Effusion=No: LTE Week 24=Missing | 0 | 4 | 10 | 14
  LTE BL: Pericardial Effusion=Missing: number analyzed (Participants) | 4 | 2 | 2 | 8
  LTE BL: Pericardial Effusion=Missing: LTE Week 24=Yes | 0 | 0 | 0 | 0
  LTE BL: Pericardial Effusion=Missing: LTE Week 24=No | 0 | 1 | 0 | 1
  LTE BL: Pericardial Effusion=Missing: LTE Week 24=Missing | 4 | 1 | 2 | 7

63. Secondary Outcome: Annualized Rate of Pericarditis Recurrence in LTE Periods Based on Investigator's Assessment
Description: Annualized Recurrence Rate is defined as number of recurrences in LTE periods for all participants/Sum of participant years in LTE period for all participants. Participant years in LTE period is defined as the time from 1st dose date of LTE period to the date of End of Study, or data cutoff date, whichever is earlier. The 95% CI was calculated using an exact method with Poisson distribution.
  Pericarditis recurrence was defined as the recurrence of typical pericarditis pain associated with supportive objective evidence of pericarditis. At any time during the RW period, participants who experienced a suspected recurrence of pericarditis symptoms reported to the study site/clinic for a scheduled or unscheduled visit, during which clinical assessments were performed to gather all the necessary diagnostic data to confirm or rule out the presence of pericarditis recurrence.
Time Frame: LTE Period, through LTE Follow up (up to Week 48)
Population: LTE Analysis Set: participants who consented to LTE period and took at least 1 dose of study drug in the LTE period.
Measure: Number (95% Confidence Interval); unit: recurrences per participant per year
Arm/Group | Long Term Extension: Non-Randomized | Long Term Extension: Randomized, Recurrence (RW) | Long Term Extension: Randomized, No Recurrence (RW) | Long-Term Extension: Overall
Number analyzed (Participants) | 15 | 25 | 34 | 74
recurrences per participant per year | 0.088 [0.011 to 0.319] | 0.168 [0.062 to 0.367] | 0.125 [0.046 to 0.273] | 0.132 [0.072 to 0.221]

64. Secondary Outcome: Annualized Rate of Pericarditis Recurrence in RW Period Based on CEC Adjudication
Description: Annualized Recurrence Rate is defined as the number of recurrences in RW period for all participants/Sum of participant years in RW period for all participants. Participant years in RW period is defined as the time from randomization date to the date of EORW or last dose date + 6 weeks, whichever is earlier. The 95% CI was calculated using an exact method with Poisson distribution.
  Pericarditis recurrence was defined as the recurrence of typical pericarditis pain associated with supportive objective evidence of pericarditis. At any time during the RW period, participants who experienced a suspected recurrence of pericarditis symptoms reported to the study site/clinic for a scheduled or unscheduled visit, during which clinical assessments were performed to gather all the necessary diagnostic data to confirm or rule out the presence of pericarditis recurrence.
Time Frame: RW Period (mean 24.8 weeks)
Population: ITT Analysis Set: all participants who were randomized in the RW period. Participants who received rilonacept in the RW period only.
Measure: Number (95% Confidence Interval); unit: recurrences per participant per year
Groups:
- Randomized Withdrawal Period: Rilonacept: Double-blind rilonacept 160 mg (or 2.2 mg/kg in pediatric participants ≥ 12 and < 18 years old) SC injections once weekly.
  Participants with pericarditis recurrence who meet the protocol criteria for bailout rilonacept (report at least 1 day with pericarditis pain ≥4 on the 11-point numerical rating scale (NRS) and have 1 C-reactive protein (CRP) value ≥ 1 mg/dL [either on the same day or separated by no more than 7 days]) receive bailout rilonacept (2 open-label injections of 160 mg rilonacept [or 4.4 mg/kg for pediatric participants]) irrespective of randomized treatment assignment and as soon as at least 5 days have passed since the last study drug injection.
Arm/Group | Randomized Withdrawal Period: Rilonacept
Number analyzed (Participants) | 30
recurrences per participant per year | 0.137 [0.017 to 0.494]

ADVERSE EVENTS:
Time Frame: All Cause Mortality: From enrollment through end of study; up to 156 weeks. Adverse events (AEs), RI Period: from first dose of study drug to the RW period randomization visit; mean duration 11.61 weeks. AEs, RW Period Rilonacept Only, Before Bailout: from RW period randomization until bailout rilonacept administration; mean duration 24.40 weeks. AEs, RW Period Rilonacept, Including Bailout Rilonacept: from RW period randomization until LTE rilonacept administration; mean duration 25.07 weeks.
Description: AEs, RW Period Placebo Only, Before Bailout: from RW period randomization to placebo until bailout rilonacept administration; mean duration was 9.88 weeks. RW Period Placebo, Including Bailout Rilonacept: from RW period randomization until LTE rilonacept administration; mean duration was 23.88 weeks. LTE period: from first dose in the LTE period until 6 weeks post last dose; mean treatment duration was 68.13 weeks. Per statistical analysis plan, safety in LTE period was reported overall only.
Groups:
- Run-in Period: Single-blind rilonacept 320 mg (or 4.4 mg/kg in pediatric participants ≥ 12 and < 18 years old) subcutaneous (SC), followed by 160 mg (or 2.2 mg/kg in pediatric subjects ≥12 and <18 years old) injections once weekly for 12 weeks.
- Randomized Withdrawal Period: Rilonacept Only, Before Bailout Rilonacept: Double-blind rilonacept 160 mg (or 2.2 mg/kg in pediatric participants ≥ 12 and < 18 years old) SC injections once weekly.
- Randomized Withdrawal Period: Placebo Only, Before Bailout Rilonacept: Double-blind placebo SC injections once weekly.
- Long-Term Extension Period: Overall: Participants received up to 24 months of open-label rilonacept 160 mg (or 2.2 mg/kg for pediatric participants) SC injections once weekly based on their clinical status and at the discretion of the Investigator.
Arm/Group | Run-in Period | Randomized Withdrawal Period: Rilonacept Only, Before Bailout Rilonacept | Randomized Withdrawal Period: Rilonacept, Including Bailout Rilonacept | Randomized Withdrawal Period: Placebo Only, Before Bailout Rilonacept | Randomized Withdrawal Period: Placebo, Including Bailout Rilonacept | Long-Term Extension Period: Overall
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/30 | 0/30 | 0/31 | 0/31 | 0/74
Serious Adverse Events (participants affected / at risk) | 1/86 | 1/30 | 1/30 | 1/31 | 3/31 | 6/74
Other Adverse Events (participants affected / at risk) | 55/86 | 18/30 | 18/30 | 7/31 | 13/31 | 43/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Period (N=86) | Randomized Withdrawal Period: Rilonacept Only, Before Bailout Rilonacept (N=30) | Randomized Withdrawal Period: Rilonacept, Including Bailout Rilonacept (N=30) | Randomized Withdrawal Period: Placebo Only, Before Bailout Rilonacept (N=31) | Randomized Withdrawal Period: Placebo, Including Bailout Rilonacept (N=31) | Long-Term Extension Period: Overall (N=74)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Aortic valve disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Acute endocarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Device malfunction (Product Issues) | 0 | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Period (N=86) | Randomized Withdrawal Period: Rilonacept Only, Before Bailout Rilonacept (N=30) | Randomized Withdrawal Period: Rilonacept, Including Bailout Rilonacept (N=30) | Randomized Withdrawal Period: Placebo Only, Before Bailout Rilonacept (N=31) | Randomized Withdrawal Period: Placebo, Including Bailout Rilonacept (N=31) | Long-Term Extension Period: Overall (N=74)
Diarrhoea (Gastrointestinal disorders) | 5 | 0 | 0 | 0 | 0 | 4
Fatigue (General disorders) | 2 | 2 | 2 | 0 | 1 | 3
Injection site erythema (General disorders) | 18 | 6 | 7 | 0 | 1 | 3
Injection site pruritus (General disorders) | 5 | 4 | 5 | 0 | 1 | 0
Injection site swelling (General disorders) | 5 | 1 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 3 | 3 | 1 | 1 | 4
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 4
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 10
Influenza (Infections and infestations) | 1 | 0 | 0 | 1 | 2 | 0
Nasopharyngitis (Infections and infestations) | 6 | 2 | 2 | 0 | 0 | 5
Sinusitis (Infections and infestations) | 1 | 3 | 3 | 0 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 3 | 3 | 0 | 1 | 5
Blood Cholesterol Increased (Investigations) | 1 | 2 | 2 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 2 | 2 | 0 | 0 | 3
High density lipoprotein increased (Investigations) | 0 | 3 | 3 | 0 | 0 | 1
Lipids increased (Investigations) | 0 | 2 | 2 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 1 | 1 | 0 | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 1 | 2 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 4 | 4 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 1 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 7 | 0 | 0 | 0 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 1 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3 | 0 | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 0 | 0 | 1
Hypertension (Vascular disorders) | 2 | 1 | 1 | 1 | 1 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the first right to publish information obtained from the trial. After sponsor publishes, PI may publish its own trial results, provided that sponsor may embargo such publication for up to 60 days for purposes of identifying confidential information (other than trial data) that must be removed and up to an additional 120 days to prepare a patent application if there is patentable subject matter in the PI's proposed publication.

DOCUMENTS (2):
  • Study Protocol (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/10/NCT03737110/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/10/NCT03737110/SAP_002.pdf